## Clinical Protocol I8B-MC-ITRM (a)

A Prospective, Randomized, Double-Blind Comparison of LY900014 to Insulin Lispro With an Open-Label Postprandial LY900014 Treatment Group, in Combination With Insulin Glargine or Insulin Degludec, in Adults With Type 1 Diabetes PRONTO-T1D

NCT03214367

Approval Date: 22-May-2017

# Clinical Protocol I8B-MC-ITRM (a) A Prospective, Randomized, Double-Blind Comparison of LY900014 to Insulin Lispro with an Open-Label Postprandial LY900014 Treatment Group, in Combination with Insulin Glargine or Insulin Degludec, in Adults with Type 1 Diabetes PRONTO-T1D

[EudraCT number: 2015-005356-99]

## **Confidential Information**

The information contained in this document is confidential and is intended for the use of clinical investigators. It is the property of Eli Lilly and Company or its subsidiaries and should not be copied by or distributed to persons not involved in the clinical investigation of LY900014, unless such persons are bound by a confidentiality agreement with Eli Lilly and Company or its subsidiaries.

Note to Regulatory Authorities: This document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

#### LY900014

Study I8B-MC-ITRM is a Phase 3, prospective, randomized, double-blind, outpatient, multinational, multicenter, 3-treatment group, parallel, active-controlled study conducted in patients with type 1 diabetes currently using a multiple daily injection regimen.

Eli Lilly and Company Indianapolis, Indiana USA 46285

Protocol Electronically Signed and Approved by Lilly: 16 Feb 2017
Amendment (a) Electronically Signed and Approved by Lilly
on approval date provided below.

Approval Date: 22-May-2017 GMT

# **Table of Contents**

| Section | Page |
|-----------------------------------------------------------------|------|
| 1. Synopsis | 8 |
| 2. Schedule of Activities | 13 |
| 3. Introduction | 20 |
| 3.1. Study Rationale | 20 |
| 3.2. Background | 20 |
| 3.3. Benefit/Risk Assessment | 22 |
| 4. Objectives and Endpoints | 23 |
| 5. Study Design | 26 |
| 5.1. Overall Design | 26 |
| 5.2. Number of Participants | 28 |
| 5.3. End of Study Definition | 28 |
| 5.3.1. Safety Follow-Up | 28 |
| 5.4. Scientific Rationale for Study Design | 28 |
| 5.5. Justification for Dose | 29 |
| 6. Study Population. | 30 |
| 6.1. Inclusion Criteria. | 30 |
| 6.2. Exclusion Criteria | 32 |
| 6.3. Lifestyle Restrictions. | 34 |
| 6.4. Screen Failures | 35 |
| 7. Treatments | 36 |
| 7.1. Treatments Administered | 36 |
| 7.1.1. Packaging and Labeling | 36 |
| 7.1.2. Medical Devices | 37 |
| 7.2. Method of Treatment Assignment | 37 |
| 7.2.1. Selection and Timing of Doses | |
| 7.2.1.1. Target Glucose Values for Titration of Insulin Therapy | |
| 7.2.1.2. Basal Insulin Therapy | |
| 7.2.1.3. Basal Insulin Titration | |
| 7.2.1.4. Study Prandial Insulin Therapy | |
| 7.2.1.5. Transitioning off Study Prandial Insulin Therapy | |
| 7.3. Blinding | |
| 7.4. Dosage Modification | |
| 7.5. Preparation/Handling/Storage/Accountability | |
| 7.6. Treatment Compliance | 43 |

| 7.7. C | oncomitant Therapy | 44 |
|----------|----------------------------------------------------|----|
| 7.8. Ti | reatment after the End of the Study | 44 |
| 7.8.1. | Continued Access | 44 |
| 7.8.2. | Special Treatment Considerations | 44 |
| 8. Disco | ontinuation Criteria | 45 |
| 8.1. D | iscontinuation from Study Treatment | 45 |
| 8.1.1. | Permanent Discontinuation from Study Treatment | 45 |
| 8.1.2. | Temporary Discontinuation from Study Treatment | 46 |
| 8.1.3. | Discontinuation of Inadvertently Enrolled Patients | 46 |
| 8.2. D | iscontinuation from the Study | 46 |
| 8.3. Lo | ost to Follow-Up | 47 |
| 9. Study | y Assessments and Procedures | 48 |
| 9.1. Et | fficacy Assessments | 48 |
| 9.1.1. | Primary Efficacy Assessments | 48 |
| 9.1.2. | Secondary Efficacy Assessments | 48 |
| 9.1.3. | Appropriateness of Assessments | 49 |
| 9.1.4. | Study Procedures | 49 |
| 9.1.4 | Electronic Clinical Outcomes Assessment | 49 |
| 9.1.4 | 2. Four-Point Self-Monitoring Blood Glucose | 49 |
| 9.1.4 | -3. Ten-Point Self-Monitoring Blood Glucose | 50 |
| 9.1.4 | .4. Mixed-Meal Tolerance Test | 50 |
| 9.1.4 | 2.5. Diabetes Education and Nutritional Counseling | 52 |
| 9.2. A | dverse Events | 52 |
| 9.2.1. | Serious Adverse Events | 53 |
| 9.2.1 | .1. Suspected Unexpected Serious Adverse Reactions | 54 |
| 9.2.2. | Complaint Handling | 54 |
| 9.3. Ti | reatment of Overdose | 54 |
| 9.4. Sa | afety | |
| 9.4.1. | Hypoglycemia | 55 |
| 9.4.2. | Severe Hypoglycemia | |
| 9.4.3. | Electrocardiograms | 56 |
| 9.4.4. | Vital Signs | |
| 9.4.5. | Laboratory Tests | |
| 9.4.6. | Safety Monitoring | |
| | narmacokinetics | |
| | narmacodynamics | |
| | narmacogenomics | |
| 9.7.1. | Whole Blood Samples for Pharmacogenetic Research | 57 |

| 9.8. Biomarkers and Predictive or Other Analyses | 57 |
|----------------------------------------------------------|----|
| 9.8.1. Samples for Immunogenicity Testing | |
| 9.9. Health Economics | |
| CCI | 56 |
| 9.9.2. Insulin Treatment Satisfaction Questionnaire | 59 |
| COL | |
| 10. Statistical Considerations | 61 |
| 10.1. Sample Size Determination | 61 |
| 10.2. Populations for Analyses | 61 |
| 10.3. Statistical Analyses | 61 |
| 10.3.1. General Statistical Considerations | 61 |
| 10.3.2. Treatment Group Comparability | |
| 10.3.2.1. Patient Disposition | |
| 10.3.2.2. Patient Characteristics | |
| 10.3.2.3. Concomitant Therapy | |
| 10.3.2.4. Treatment Compliance | 64 |
| 10.3.3. Efficacy Analyses | |
| 10.3.3.1. Primary Analyses | |
| 10.3.3.1.1. Sensitivity Analyses for Missing Data | |
| 10.3.3.1.2. Additional Analyses for the Primary Endpoint | |
| 10.3.3.2. Secondary Analyses | |
| 10.3.3.3. Tertiary/Exploratory Analyses | |
| 10.3.4. Safety Analyses | |
| 10.3.5. Other Analyses | |
| 10.3.5.1. Health Economics | 68 |
| 10.3.5.2. Subgroup Analyses | |
| 10.3.6. Interim Analyses | |
| 11. References | |
| 12. Appendices | |
| - Production | |

## **List of Tables**

| Table | | Page |
|---|---|---|
| Table ITRM.1. | Objectives and Endpoints | 23 |
| Table ITRM.2. | Treatment Regimens | 36 |
| Table ITRM.3. | Target Glucose Values for Adjustment of Insulin Therapy | 37 |
| Table ITRM.4. | Basal Insulin Hypoglycemia Assessment | 39 |
| Table ITRM.5. | Summary of Basal Insulin Adjustments after Hypoglycemia Assessment | 39 |
| Table ITRM.6. | Prandial Insulin Doses and Corresponding Self Monitored Blood<br>Glucose Values Pattern Adjustment Plan | 41 |
| Table ITRM.7. | LY900014 or Insulin Lispro Adjustment Algorithm Pattern Adjustment Plan | 42 |
| Table ITRM.8. | Concomitant Medications | 44 |
| Table ITRM.9. | Insulin to Carbohydrate Ratio for Determining the Prandial Insulin dose for the Mixed-Meal Tolerance Test: For Use with Patients who use Pattern Adjustment to Determine Prandial Insulin Doses | 51 |
| Table ITRM.10. | Summary of Basal Insulin Adjustments after Hypoglycemia Assessment | 99 |

| Ρ | a | a | е | 6 |
|---|---|---|---|---|

| Li | st ( | of | Fig | jures | , |
|----|------|----|-----|-------|---|

| Figure | • | Page |
|---|---|---|
| Figure ITRM.1. | Illustration of study design for Clinical Protocol I8B-MC-ITRM | 27 |

# **List of Appendices**

| Appendix | | Page |
|---|---|---|
| Appendix 1. | Abbreviations and Definitions | 74 |
| Appendix 2. | Clinical Laboratory Tests | 78 |
| Appendix 3. | Study Governance Considerations | 79 |
| Appendix 4. | Hepatic Monitoring Tests for Treatment-Emergent Abnormality | 83 |
| CCI | | |
| Appendix 6. | New York Heart Association Cardiac Disease Classification | 85 |
| Appendix 7. | Classification of Contraceptive Methods | 86 |
| Appendix 8. | Insulin Lispro Antibody Follow-Up Assessment | 87 |
| Appendix 9. | Protocol Amendment I8B-MC-ITRM(a) Summary A Prospective,<br>Randomized, Double-Blind Comparison of LY900014 to Insulin Lispro<br>with an Open-Label Postprandial LY900014 Treatment Group, in<br>Combination with Insulin Glargine or Insulin Degludec, in Adults with<br>Type 1 Diabetes | |
| | PRONTO-T1D | 91 |

# 1. Synopsis

#### Title of Study:

A Prospective, Randomized, Double-Blind Comparison of LY900014 to Insulin Lispro with an Open-Label Postprandial LY900014 Treatment Group, in Combination with Insulin Glargine or Insulin Degludec, in Adults with Type 1 Diabetes PRONTO-T1D

#### **Rationale:**

Prandial insulin with faster-onset and/or faster-offset characteristics might reduce glycemic excursions and the incidence of delayed postprandial hypoglycemia compared to currently available rapid-acting insulin analogs. Rapid-acting insulins, such as Humalog®, have been shown to have a more rapid onset of action compared to human insulin; however, the general consensus is that they are not rapid enough to match carbohydrate absorption, whether delivered by pump or syringe/pen injector, limiting efficacy. An ultra-rapid-acting prandial insulin that would shift the pharmacokinetic (PK) and glucodynamic profiles of insulin to provide an even faster onset of action would better match carbohydrate absorption and allow for efficacious dosing immediately prior to meals or even after meals. Ultra-rapid insulin (URI) could be useful in the treatment of type 1 diabetes (T1D) and type 2 diabetes (T2D) in adults and children when given by multiple daily injections (MDI) or by continuous subcutaneous insulin infusion (CSII).

The aim of this study is to demonstrate that an ultra-rapid formulation of insulin lispro, LY900014, is noninferior to insulin lispro on glycemic control as measured by change from baseline to Week 26 in hemoglobin A1c (HbA1c) in patients with T1D when administered in a double-blind manner as prandial insulin in combination with basal insulin glargine or insulin degludec.

## **Objectives/Endpoints:**

Note: Week 52 endpoints for the secondary objectives only apply to the blinded treatment arms of LY900014 and insulin lispro.

| Objectives | Endpoints |
|---|---|
| Primary Objective | |
| 1. To test the hypothesis that LY900014 is noninferior to insulin lispro on glycemic control (noninferiority margin [NIM]=0.4% for hemoglobin A1c [HbA1c]) in patients with T1D, when administered as prandial insulin (0 to 2 minutes prior to the meal), in combination with basal insulin glargine or insulin degludec for 26 weeks | Difference between LY900014 and insulin lispro in change from baseline to Week 26 in HbA1c |
| <b>Multiplicity Adjusted Objectives</b> | |
| 2. To test the hypothesis that LY900014 is superior to insulin lispro in controlling 1-hour postprandia glucose (PPG) excursions, when administered as prandial insulin | 2. Difference between LY900014 and insulin lispro in the 1-hour PPG excursion (serum glucose measured 1 hour after the start of the meal minus fasting serum glucose) from a mixed-meal tolerance test (MMTT) at Week 26 |

| 3. | To test the hypothesis that LY900014 is superior | 3. Difference between LY900014 and ins | sulin lispro |
|---|---|---|---|
| σ. | to insulin lispro in controlling 2-hour PPG excursions, when administered as prandial insulin | in the 2-hour PPG excursion (serum gl<br>measured 2 hours after the start of the<br>fasting serum glucose) from an MMTT | ucose<br>meal minu |
| | | Week 26 | . at |
| 4. | To test the hypothesis that LY900014 is superior to insulin lispro on improving glycemic control (HbA1c) when administered as prandial insulin | 4. Difference between LY900014 and ins in change from baseline to Week 26 in | - |
| 5. | To test the hypothesis that LY900014 administered as postprandial insulin 20 minutes after the start of a meal (LY900014+20), is noninferior to insulin lispro, administered as prandial insulin, on glycemic control (NIM=0.4% for HbA1c) | 5. Difference between LY900014+20 and lispro in change from baseline to Weel HbA1c | |
| Othe | r Secondary Objectives | | |
| 6. | To compare LY900014+20 with insulin lispro and LY900014 with respect to 1-hour and 2-hour PPG excursions | 6. 1- and 2-hour PPG excursions from an Week 26 | MMTT at |
| 7. | To compare the glycemic control of LY900014 with LY900014+20 | 7. Change from baseline HbA1c values a | t Week 26 |
| 8. | To compare LY900014, LY900014+20, and insulin lispro on the rate of severe hypoglycemic events | 8. Rate (events/patient/100 years) of seven hypoglycemic events from baseline thrule Week 26 and Week 52 | |
| 9. | To compare LY900014, LY900014+20, and insulin lispro with respect to the incidence and rate of documented symptomatic postmeal hypoglycemia | 9. Rate (events/patient/year and/or events/patient/30 days) and incidence (patients with at least 1 event) of docum symptomatic postmeal hypoglycemia v 2 hours after start of a meal from Weel through Week 26, Week 0 through Week 26 through Week 52, and Week Week 52 | nented<br>within 1 an<br>k 12<br>eek 26, |
| 10. | To compare LY900014, LY900014+20, and insulin lispro with respect to the incidence and rate of documented symptomatic hypoglycemia | 10. Rate (events/patient/year and/or events/patient/30 days) and incidence (patients with events) of documented sy hypoglycemic events from Week 12 th Week 26, Week 0 through Week 26, W through Week 52, and Week 0 through | ymptomation<br>rough<br>Veek 26 |
| 11. | To compare LY900014, LY900014+20, and insulin lispro with respect to 1,5-Anhydroglucitol (1,5-AG) | 11. Change from baseline 1,5-AG values a and Week 52 | nt Week 26 |
| 12. | To compare LY900014, LY900014+20, and insulin lispro with respect to 10-point self-monitored blood glucose (SMBG) profiles | 12. Change from baseline 10-point SMBG Week 26 and Week 52 | values at |
| 13. | To compare LY900014, LY900014+20, and insulin lispro with respect to total, basal, and prandial insulin dose | 13. Change from baseline in total, basal an insulin doses and prandial/total insulin at Week 26 and Week 52 | • |

| 14. To compare LY900014, LY900014+20, and insulin lispro with respect to diabetes treatment satisfaction as measured by the Insulin Treatment Satisfaction Questionnaire (ITSQ) | 14. Change from baseline in ITSQ regimen inconvenience and lifestyle flexibility domain scores at Week 26 and Week 52 |
|---|---|
| 15. To compare LY900014, LY900014+20, and insulin lispro with respect to the proportion of patients achieving HbA1c targets | 15. The proportion of patients with HbA1c <7% and ≤6.5% at Week 26 and Week 52 |
| To compare the glycemic control of LY900014 and insulin lispro | 16. Actual and change from baseline to Week 52 in HbA1c |

#### **Summary of Study Design:**

Study I8B-MC-ITRM is a Phase 3, prospective, randomized, double-blind, outpatient, multinational, multicenter 3-treatment group, parallel, active-controlled study in patients with T1D currently using an MDI regimen.

### **Treatment Groups and Duration:**

The study includes a 1-week screening period and an 8-week lead-in period. In 2 of the treatment groups, LY900014 and insulin lispro will be administered immediately (0-2 minutes) prior to each meal in a double-blind manner. Patients in these groups will complete a 52-week treatment period (with primary endpoint at 26 weeks), and a 4-week safety follow-up period. A third open-label treatment group consists of LY900014 administered 20 minutes after the start of a meal (LY900014+20). Patients in this treatment group will complete a 26-week treatment period and the 4-week safety follow-up period.

All patients who complete the 4-week safety follow-up visit (Visit 801) and have treatment-emergent insulin lispro antibodies that have not returned to prespecified baseline range (Visit 2) will be asked to participate in follow-up to monitor insulin lispro antibody levels. Study visits will be scheduled at approximately 3-month intervals for up to 26 weeks from Visit 801 or until insulin lispro antibodies return to baseline range, whichever occurs sooner.

#### **Number of Patients:**

Approximately 1500 participants will be screened to achieve 1199 randomized patients and 1020 patients completing 26 weeks of treatment, with approximately 646 patients completing 52 weeks.

## **Statistical Analysis:**

The primary analysis is for the treatment period through Week 26.

Efficacy analyses will be conducted on all randomized patients according to the treatment the patients are assigned. The analyses for the primary and multiplicity adjusted objectives will be performed for the efficacy estimand including data collected prior to permanent discontinuation of investigational product (IP) through Week 26 and for the ITT estimand (treatment regimen estimand) including all data collected through Week 26 regardless of IP use. When change from baseline is included as a response variable of analysis models, the patient will be included in the analysis only if a baseline and at least 1 postbaseline measurement are available. Selected efficacy analyses will also be conducted using the Per Protocol (PP) and Completer populations. Week 52 analyses will include the LY900014 and insulin lispro treatment arms and only be performed for the efficacy estimand.

Safety analyses will be conducted on the Safety population. Analyses of adverse events (AEs) will include 2 sets of analyses, unless otherwise specified. The first set of analyses will include data collected prior to permanent

discontinuation of IP. The second set of analyses will include all data collected during the course of the entire study regardless of IP use. Analyses of hypoglycemia will be conducted on data collected prior to permanent discontinuation of IP, while analyses for post-treatment may be conducted as needed. Analyses of safety laboratory measurements will be performed on all data collected during the planned treatment period regardless of IP use. Week 26 analyses will include treatment comparisons among three treatment groups. Week 52 analyses will also include data collected during the follow-up visit for LY900014 and insulin lispro. All data collected including the follow-up visit will be summarized for LY900014+20.

Baseline is defined as the last nonmissing measurement at or before the randomization visit (Visit 8), unless otherwise specified.

For the US Food and Drug Administration (FDA) submission, the primary analysis method will use the copy reference approach to impute missing data based on multiple imputations with a pattern mixture model. This analysis is for the ITT estimand that will include all data collected from randomization through Week 26, regardless of IP use. The reference will be all observed data from the randomized patients in the same treatment arm who discontinue IP and complete the study without missing data. After imputation, the primary efficacy comparison will be based on the contrast between LY900014 and insulin lispro from the analysis of covariance (ANCOVA) analysis of change from baseline to Week 26 in HbA1c using all randomized patients. The model for this analysis will include the fixed class effects of treatment and strata (pooled country, type of basal insulin, and prandial insulin dosing plan), and the continuous, fixed covariate of baseline value.

If there are only a limited number of patients in the reference group as described above that leads to a failure in performing the proposed multiple imputation analysis, the reference will be changed to include all observed data from all randomized patients in the same treatment arm who complete the study without missing data.

For non-FDA submissions and publications, the primary efficacy comparison will be based on the contrast between LY900014 and insulin lispro at Week 26 (Visit 18) from the mixed-effect model repeated measure (MMRM) analysis of change from baseline in HbA1c including data collected from all randomized patients prior to permanent discontinuation of IP through Week 26 (efficacy estimand). The model for this analysis will include the fixed class effects of treatment and strata (pooled country, type of basal insulin, and prandial insulin dosing plan), visit, and treatment-by-visit interaction, and the continuous, fixed covariate of baseline value.

For both primary analysis approaches, LY900014 will be declared noninferior to insulin lispro if the upper limit of the 2-sided 95% confidence interval (CI) for the least squares (LS) mean difference in the change from baseline in HbA1c for LY900014 minus insulin lispro is below +0.4%. In addition, the 95% CI for the treatment difference will be compared to an alternative NIM of +0.3%. Both estimands will be tested at the full significance level of 0.05. The ANCOVA and MMRM analyses will include data from all 3 treatment groups; however, the contrasts between LY900014+20 and insulin lispro and between LY900014 and LY900014+20 are not part of the primary efficacy comparisons.

A graphical approach (Bretz et al. 2011) for multiple comparisons will be used to strongly control the overall Type I error (2-sided alpha level of 0.05) for testing the treatment effect for the primary and the following multiplicity adjusted objectives: superiority of LY900014 compared with insulin lispro for 1-hour PPG excursion at Week 26, 2-hour PPG excursion at Week 26, and change from baseline to Week 26 in HbA1c; and noninferiority of LY900014+20 to insulin lispro in change from baseline to Week 26 in HbA1c. The same graphical testing scheme will be applied for both the efficacy estimand and ITT estimand.

An analysis of covariance (ANCOVA) model with strata (pooled country, type of basal insulin, baseline HbA1c strata [(≤7.5%, >7.5%], and prandial insulin dosing plan during the study), and treatment as fixed effects and baseline as a covariate will be used to analyze the 1-hour and 2-hour PPG excursions. However, if the percentage of the patients with missing MMTT data at baseline is higher than 15%, a constrained longitudinal data analysis model (Liu et al. 2009; Lu 2010) will be used instead. Analyses details will be documented in the statistical analysis plan (SAP).

Hypoglycemia rates will be summarized for periods of 30 days, 1 year, and 100 years (severe hypoglycemia only). The rate of severe hypoglycemia per 100 years will be compared between treatment groups using the empirical method. For each of the other categories of hypoglycemia, the number of hypoglycemia events during a specific period (rate) after randomization (for example, 0-12 weeks of treatment period) will be analyzed by using a negative binomial regression model. The model will include treatment and the baseline hypoglycemia rate (measured during lead-in) as a covariate. An offset defined as the log transformation of treatment exposure in the specific period (days)/365.25 days (or 30 days) will be included in the model to estimate the rate of hypoglycemia per year (or per 30 days). The proportion of patients with at least 1 hypoglycemic event in each category (incidence) during a specific period after randomization will be analyzed using a logistic regression model including treatment and baseline hypoglycemia rate value in the model.

Continuous safety variables, as well as the change from baseline for these variables, will be analyzed by MMRM or ANCOVA models. For categorical variables, Fisher's exact test or Pearson's chi-square test will be used to compare treatment groups unless otherwise specified.

Change from baseline to last-observation-carried forward endpoints for the CCI

ITSQ, and CCI

will be analyzed using ANCOVA models.

#### References:

Bretz F, Posch M, Glimm E, Klinglmueller F, Maurer W, Rohmeyer K. Graphical approaches for multiple comparison procedures using weighted Bonferroni, Simes, or parametric tests. Biom J. 2011;53(6):894-913.

Liu GF, Lu K, Mogg R, Mallick M, Mehrotra DV. Should baseline be a covariate or dependent variable in analyses of change from baseline in clinical trials? Stat Med. 2009;28(20):2509-2530.

Lu K. On efficiency of constrained longitudinal data analysis versus longitudinal analysis of covariance. Biometrics. 2010;66(3):891-896.

# 2. Schedule of Activities

| Study Procedure | Study<br>Screening | | L | ead-I | n Per | riod | | | Ir | ntensi | ve Titi<br>Prim | ration | | | Perio | | Maintenance<br>Period | | | ntena<br>uble B | Term nce Pe | eriod | Safety<br>Follow-<br>Up | ED |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| eCRF Visit Number | 1 | 2 | 3a | 4a | 5 | 6a | 7 | 8 | 9a | 10 | 11 | 12<br>a | 13 | 14<br>a | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 801 | EDp |
| Visit Window<br>(± days) | | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | |
| Time on Study Relative to First Active Treatment Dose (weeks) | -9 | -8 | -7 | -6 | -4 | -2 | -1 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 18 | 22 | 26 | 32 | 39 | 46 | 52 | 56 (30) <sup>c</sup> | |
| Informed consent signed | X | | | | | | | | | | | | | | | | | | | | | | | |
| IWRS | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Patient eligibility review | X | | | | | | | | | | | | | | | | | | | | | | | |
| Randomizationd | | | | | | | | X | | | | | | | | | | | | | | | | |
| Telephone call for<br>visit reminder or<br>informing patient of<br>completion in the<br>study | | | | | | | | | | | | | | | | | | | | | | | X | |
| Clinical Assessments | | | | | | | l | ı | | | I | | | | | ı | ı | I | 1 | I | I | 1 | | |
| Patient demographics | X | | | | | | | | | | | | | | | | | | | | | | | |
| Medical history and preexisting conditions | X | | | | | | | | | | | | | | | | | | | | | | | |
| Physical exam/height | X | | | | | | | | | | | | | | | | | | | | | | | |
| Concomitant medication | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events and product complaints | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

| Study Procedure | Study<br>Screening | | L | ead-I | n Per | riod | | | Iı | ntensi | ve Titi<br>Prim | ration<br>nary T | | nce<br>I | Mai | Long<br>ntenai<br>ible B<br>On | nce Po | Safety<br>Follow-<br>Up | ED | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| eCRF Visit Number | 1 | 2 | 3a | 4a | 5 | 6a | 7 | 8 | 9a | 10 | 11 | 12<br>a | 13 | 14<br>a | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 801 | EDp |
| Visit Window<br>(± days) | | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | |
| Time on Study Relative to First Active Treatment Dose (weeks) | -9 | -8 | -7 | -6 | -4 | -2 | -1 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 18 | 22 | 26 | 32 | 39 | 46 | 52 | 56 (30) <sup>c</sup> | |
| Body weighte | X | X | | | X | | X | X | | X | X | | X | | X | X | X | X | X | X | X | X | X | X |
| Vital signs: blood<br>pressure/pulse ratef | X | X | | | X | | X | X | | X | X | | X | | X | X | X | X | X | X | X | X | X | X |
| ECG <sup>g</sup> (12-lead; local) | X | | | | | | | | | | | | | | | | | | | | | | | |
| Diabetes and nutrition counselingh | | X | | | | | | | | | | | | | | | | | | | | | | |
| Transfer to insulin lisproi | | X | | | | | | | | | | | | | | | | | | | | | | |
| Transfer to allowed study basal insulin regimeni | | X | | | | | | | | | | | | | | | | | | | | | | |
| Basal and prandial insulin dose assessment <sup>k</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Titrate basal insulink | | X | X | X | X | X | X | | | | | | | | | | | | | | | | | |
| Titrate prandial insulin <sup>1</sup> | | | | | | | | X | X | X | X | X | X | X | X | | | | | | | | | |

| <b>Study Procedure</b> | Study<br>Screening | | Le | ead-I | n Pei | riod | | | Ir | itensi | ve Titi | | | | | | intena<br>Perioc | | Mai | Long<br>ntena | nce Po | eriod | Safety<br>Follow- | ED |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | Prin | nary T | reati | ment ] | Perio | d | | | (Doi | uble B<br>Or | Blind A<br>nly) | Arms | Up | |
| eCRF Visit Number | 1 | 2 | 3a | 4a | 5 | 6a | 7 | 8 | 9a | 10 | 11 | 12<br>a | 13 | 14<br>a | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 801 | EDp |
| Visit Window | | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | |
| (± days) | | | | | | | | | | | | | | | | | | | | | | | | |
| Time on Study | -9 | -8 | -7 | -6 | -4 | -2 | -1 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 18 | 22 | 26 | 32 | 39 | 46 | 52 | 56 (30) <sup>c</sup> | |
| Relative to First | | | | | | | | | | | | | | | | | | | | | | | ` ' | |
| <b>Active Treatment</b> | | | | | | | | | | | | | | | | | | | | | | | | |
| Dose (weeks) | | | | | | | | | | | | | | | | | | | | | | | | |
| Ancillary Supplies/Di | aries/IP | | | | | | | | | | | | | | | | | | | | | | | |
| Dispense blood | | X | | | | | | X | | X | X | | X | | X | X | X | X | X | X | X | X | X | |
| glucose meter and | | | | | | | | | | | | | | | | | | | | | | | | |
| ancillary supplies and | | | | | | | | | | | | | | | | | | | | | | | | |
| complete training <sup>m,n</sup> | | | | | | | | | | | | | | | | | | | | | | | | |
| Dispense eCOA and | | X | | | | | | | | | | | | | | | | | | | | | | |
| complete training <sup>n</sup> | | | | | | | | | | | | | | | | | | | | | | | | |
| Train on collecting 4- | | X | | | | | | | | | | | | | | | | | | | | | | |
| and 10-point SMBG | | | | | | | | | | | | | | | | | | | | | | | | |
| profiles <sup>n</sup> | | | | | | | | | | | | | | | | | | | | | | | | |
| Review 4-point | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| SMBG profiles | | | | | | | | | | | | | | | | | | | | | | | | |
| Remind patient of 10- | | | | | | X | X | | | X | | X | | X | | | X | | X | | X | | | |
| point SMBG | | | | | | | | | | | | | | | | | | | | | | | | |
| requirementso | | | | | | | | | | | | | | | | | | | | | | | | |
| Review 10-point | | | | | | | | X | | | X | | X | | X | | | X | | X | | X | | Хp |
| SMBG Profiles | | | | | | | | | | | | | | | | | | | | | | | | |
| Review/discuss hypo | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| data | | | | | | | | | | | | | | | | | | | | | | | | |
| Dispense IP | | X | | | X | | | X | | | X | | X | | X | X | X | X | X | X | X | | | |
| Return of eCOA | | | | | | | | | | | | | | | | | | | | | | | X | X |
| devices | | | | | | | | | | | | | | | | | | | | | | | | |

| Study Procedure | Study<br>Screening | | Le | ead-I | n Per | riod | | | In | tensi | ve Titı | | | | | | intena<br>Period | | Mai | Long<br>ntena | nce Pe | eriod | Safety<br>Follow- | ED |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | Prim | ary T | reatr | nent l | Perio | d | | | (Dou | uble B<br>On | Blind A<br>nly) | Arms | Up | |
| eCRF Visit Number | 1 | 2 | 3a | 4a | 5 | 6a | 7 | 8 | 9a | 10 | 11 | 12<br>a | 13 | 14<br>a | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 801 | EDp |
| Visit Window<br>(± days) | | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | |
| Time on Study Relative to First Active Treatment Dose (weeks) | -9 | -8 | -7 | -6 | -4 | -2 | -1 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 18 | 22 | 26 | 32 | 39 | 46 | 52 | 56 (30) <sup>c</sup> | |
| Patient returns used<br>and unused study<br>drug supplies | | | | | X | | | X | | | X | | X | | X | X | X | X | X | X | X | X | | X |
| Drug accountability | | | | | X | | | X | | | X | | X | | X | X | X | X | X | X | X | X | | X |
| Laboratory Assessme | nts | • | • | | | | | , | | 1 | 1 | | | | | | | | | | | | | |
| Patient fasts prior to visit | | X | | | | | | X | | | | | | | | | | X | | | | X | | X |
| MMTTq | | | | | | | | X | | | | | | | | | | X | | | | | | |
| Urinalysis panel | X | | | | | | | | | | | | | | | | | | | | | | | |
| Pregnancy test <sup>r</sup> | X | | | | | | | X | | | | | | | | | | | | | | | | |
| Follicle-stimulating hormone tests | X | | | | | | | | | | | | | | | | | | | | | | | |
| Chemistry panel | X | | | | | | | X | | | | | | | | | | X | | | | X | | X |
| Fasting Serum<br>Glucose | | X | | | | | | | | | | | | | | | | | | | | | | |
| Hematology | X | | | | | | | X | | | | | | | | | | X | | | | X | | X |
| 1,5-Anhydroglucitol | | | | | | | | X | | | X | | | | X | | | X | | X | | X | | X |
| Hemoglobin A1c | X | | | | | | X | X | | | X | | X | | X | | | X | | X | | X | X | X |
| Lipid profile | | | | | | | | X | | | | | | | | | | X | | | | X | | X |
| Pharmacogenetic sample <sup>t</sup> | | | | | | | | X | | | | | | | | | | | | | | | | |

I8B-MC-ITRM Clinical Protocol Page 17

| Study Procedure | Study<br>Screening | | Le | ead-I | n Pei | riod | | | Iı | itensi | ve Titi | ration | Peri | od | | | intena<br>Period | | ı | | Term<br>nce Pe | | Safety<br>Follow- | ED |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | Prin | ary T | reatı | nent l | Perio | d | | | (Dot | | lind A<br>lly) | Arms | Up | |
| eCRF Visit Number | 1 | 2 | за | 4a | 5 | 6ª | 7 | 8 | 9a | 10 | 11 | 12<br>a | 13 | 14<br>a | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 801 | EDp |
| Visit Window<br>(± days) | | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | |
| Time on Study Relative to First Active Treatment Dose (weeks) | -9 | -8 | -7 | -6 | -4 | -2 | -1 | 0 | 1 | 2 | 4 | 6 | 8 | 10 | 12 | 18 | 22 | 26 | 32 | 39 | 46 | 52 | 56 (30) <sup>c</sup> | |
| Nonpharmacogenetic<br>biomarker storage<br>samples | | | | | | | | X | | | | | | | | | | X | | | | | | X |
| Anti-insulin lispro<br>antibodies | | X | | | | | | Х | | Х | X | | | | Х | | | X | | | | X | Xu | X |
| Health Outcomes Que | estionnairesv | | | | | | | | | | | | | | | | | | | | | | | |
| ITSQ | | Х | | | | | | X | | | | | | | | | | X | | | | X | | X |
| CCI | | X<br>X | | | | | | X | | | | | | | | | | X | | | | X | | X |

#### Schedule of Activities

Abbreviations: ECG = electrocardiogram; eCOA = electronic clinical outcomes assessment, eCRF = electronic case report form; ED = early discontinuation;

CCI

glucose; hypo = hypoglycemia; IP = investigational product; ITSQ = Insulin Treatment

Satisfaction Questionnaire; IWRS = interactive web response system; MMTT = mixed-meal tolerance test; SMBG = self-monitored blood glucose; V = visit;

- Telephone visits are indicated by shaded columns. Activities include:
  - Record visit in the IWRS.
  - Collect adverse events and concomitant medications.
  - Review blood glucose readings and study drug doses.
  - Adjust prandial insulin or basal insulin doses as needed.
  - Review hypoglycemic events.
  - Provide reminders regarding scheduled visits, fasting, and SMBG profiles, as applicable.
- Patients who have been randomized will be asked to return for the ED visit in a fasting state unless patient is already fasting and at the site when the decision to discontinue is made. Patients who discontinue during the lead-in period prior to randomization who are not already at the site, will be asked to return for the ED in a nonfasting state and all activities should be completed except for laboratory tests and questionnaires (ITSQ, CC).
- e Patients randomized to the open-label treatment group will complete the study at Week 30 unless patient continues into the insulin antibody assessment period. It is recommended that the first insulin lispro antibody follow-up visit (Visit 802 [Appendix 8]) be scheduled for all study patients, regardless of treatment-emergent antibody status. Visit 802 should occur approximately 13 weeks after Visit 801.
- d Randomization should occur after all Visit 8 procedures including MMTT. If MMTT is rescheduled post Visit 8, randomization should not occur until baseline MMTT is completed. The patient will administer their first dose of study insulin with the first meal after the MMTT has been completed and randomization has occurred.
- e Patients should be advised to remove their shoes and empty their pockets before the body weight is obtained.
- Vital sign measurements must be taken before obtaining an ECG tracing and before collection of blood samples for laboratory testing. These measurements should be determined after patients have been seated quietly for at least 5 minutes in a chair with feet on the floor. The arm used for blood pressure measurement should be supported at heart level.
- g Patients must be supine for approximately 5 to 10 minutes before ECG collection and remain supine but awake during ECG collection.
- h Initial training at Visit 2 will include diabetes education and nutrition counseling. Appropriate site personnel will administer training and education using locally approved diabetes education/training materials or other materials provided by the Sponsor. Patients may be provided abbreviated training and education at visits following Visit 2 as appropriate.
- i Only applies to patients on insulin glulisine or insulin aspart.
- Patients will be transferred to a study basal insulin regimen at Visit 2. Investigators will determine the appropriate basal insulin regimen for each patient. It is expected that most of the basal insulin dose adjustments should occur during the lead-in period. However, basal insulin titration may continue during the intensive titration period for patients who need more intensification to achieve glycemic targets. Basal insulin dose adjustments during the maintenance period should be made for safety reasons such as hypoglycemia and unacceptable hyperglycemia.
- k Assessments of the basal insulin dose should be made, at minimum, weekly during the lead-in period, including Weeks -5 and -3. Assessment of the prandial insulin dose should be made, at minimum, weekly during the initial 12 weeks after randomization, including Weeks 3, 5, 7, 9, and 11.

- During the lead-in period, prandial doses, correction factors, and insulin to carbohydrate ratios should be evaluated and adjustments should be made for safety reasons such as hypoglycemia and unacceptable hyperglycemia. During the intensive titration period, prandial insulin dose should be adjusted in order to meet the target SMBG levels. Further adjustments during the maintenance period should be made for safety reasons such as hypoglycemia and unacceptable hyperglycemia.
- m Glucose monitoring supplies will be dispensed at other visits, as needed.
- <sup>n</sup> Training may be repeated at other visits, as needed.
- o Patients in all 3 study arms should be instructed to perform three 10-point SMBG profiles during a 2-week period. The 10-point profile is completed over a 1-day period, preferably on 3 nonconsecutive days (weekdays and weekends). Ten-point SMBG profiles should not be performed on the day of MMTT.
- P Review of 10-point SMBG profiles at the ED visit will take place only for patients randomized into the study.
- 4 MMTT can occur 0 to 4 days prior to the visit, and patient must be fasting prior to start of the MMTT.
- F Serum pregnancy test must be performed in women of childbearing potential at Visit 1 followed by a urine pregnancy test within 24 hours prior to IP exposure at randomization (Visit 8) and at other times at the investigator's discretion. When required per local regulations and/or institutional guidelines, local pregnancy testing will occur at mandatory times during the study treatment period.
- s Follicle-stimulating hormone test must be performed at Visit 1 for a postmenopausal woman who is between 50 and 54 years of age (inclusive) with an intact uterus, not on hormone therapy, and who has had at least 6 months of spontaneous amenorrhea.
- t Pharmacogenetic sample can be collected at any other visit if not collected at Visit 8
- Patients with treatment-emergent insulin lispro antibodies measured at Visit 801 that have not returned to prespecified baseline range (Visit 2), will be asked to undergo additional antibody monitoring as described in Appendix 8. This follow-up assessment also applies to any patient who discontinues study insulin treatment prior to the end of the planned treatment period who has a treatment-emergent antibody response that has not returned to baseline range by Visit 801. It is recommended that the first insulin lispro antibody follow-up visit (Visit 802) be scheduled for all study patients, regardless of treatment-emergent antibody status.
- v Health outcomes questionnaires will be administered at the study sites based on the availability of appropriate translations. The questionnaires should be administered prior to other study procedures except at Visit 8 and Visit 18 when questionnaires may be administered following the start of the MMTT.

## 3. Introduction

# 3.1. Study Rationale

Prandial insulin with faster-onset and/or faster-offset characteristics might reduce glycemic excursions and decrease the incidence of delayed postprandial hypoglycemia compared to currently available rapid-acting insulin analogs. The insulin analog, insulin lispro (Humalog®), has been shown to be absorbed more quickly than regular human insulin (Humalog package insert, 2015). In healthy volunteers given subcutaneous (SC) doses of insulin lispro ranging from 0.1 to 0.4 U/kg, peak serum levels were seen 30 to 90 minutes after dosing. Rapid-acting insulins have been shown to have a more rapid onset of action compared to human insulin; however, the general consensus is that they are not rapid enough to match carbohydrate absorption and many patients are unable to achieve optimal glycemic control. An ultra-rapidacting prandial insulin with pharmacokinetic (PK) and glucodynamic (GD) profiles that demonstrate faster absorption and onset of action may better match carbohydrate absorption and lead to improved postprandial control. The time action profile of rapid-acting insulin could be enhanced through the addition of excipients to an existing formulation to increase capillary blood flow and/or enhance vascular permeability. An ultra-rapid insulin (URI) would be useful in the treatment of type 1 diabetes (T1D) and type 2 diabetes (T2D) when delivered by multiple daily injections (MDI), by continuous SC insulin infusion (CSII), and in the development of closed loop insulin delivery systems.

The aim of this study is to demonstrate that an ultra-rapid formulation of insulin lispro, LY900014, is noninferior to insulin lispro on glycemic control as measured by change from baseline to Week 26 in hemoglobin A1c (HbA1c) in patients with T1D, when administered in a double-blind manner as prandial insulin in combination with basal insulin glargine or insulin degludec.

# 3.2. Background

T1D is an autoimmune disease mediated by a combination of genetic and environmental triggers resulting in lymphocytic infiltration of pancreatic islets, destruction of beta cells, and lifelong dependency on exogenous insulin. T1D prevalence is near 1 in 300 and its incidence is steadily increasing worldwide (3% per year [Gan et al. 2012]).

There have been many advances in the treatment of T1D in the last 20 years; however, reaching and maintaining glycemic goals remains challenging even under intensive insulin therapy regimens. Only approximately 30% of insulin requiring diabetes patients are able to reach the goal HbA1c target of <7% (Stark-Casagrande et al. 2013). Currently available rapid-acting insulin analogs continue to be unable to match the kinetics of physiological postmeal insulin secretion, which is biphasic. Normal first phase insulin response is a rapid but short-lived increase in secretion, which is then followed by a more slowly developing prolonged increase (Barrett et al. 2016). First phase insulin release prevents the rapid development of postprandial hyperglycemia while second phase release of insulin ensures that glucose enters tissues in a steady, controlled manner throughout the late postprandial period. Thus, there remains a need to

continue to develop formulations with a time action profile that more closely approximates that of endogenous insulin section.

Ideally, currently available rapid-acting insulin analogs should be injected 10 to 15 minutes prior to meal consumption in order to control postprandial glucose (PPG). However, many persons inject their rapid-acting insulin at the time of the meal or after the meal. According to survey data from the T1D Exchange on the timing of prandial insulin injection, 16.3% of patients indicated that they inject 15 minutes prior to meals, 33% inject 1 to 14 minutes prior to meals, 38.6% inject at the time of the meal, and 12.1% inject after meals. Because patients often inject later than recommended there is a greater mismatch between insulin action and postprandial blood glucose (BG) elevations. With postmeal dosing, the mismatch between the rise in BG and the onset of insulin action is even more pronounced. For the development of a URI, it will be important to understand the relationship between time action profile of the insulin, insulin injection timing, and meal timing in order to maximize improvements in postprandial glycemic control and minimize hypoglycemia risk. A URI with higher early insulin concentration and peak exposure, and shorter duration should improve early postprandial control and limit postmeal hyperglycemia, while reducing late postprandial hypoglycemia due to lower insulin exposure.

HbA1c provides an integrated measurement of both fasting and postprandial glycemic control and is the most reliable marker for overall glucose exposure. Elevation in HbA1c is the best predictor of diabetes complications. Control of both fasting and postprandial hyperglycemia is essential to reach HbA1c goals. The relative contribution of postprandial hyperglycemia is predominant with moderate to fairly well controlled HbA1c levels (Monnier et al. 2003).

A new pharmaceutical innovation that may allow more effective control of PPG levels is LY900014, a new formulation of insulin lispro developed as an ultra-rapid acting insulin with a faster onset of action and shorter duration of action compared to currently available rapid-acting insulin analogs. The changes in PK and GD characteristics are achieved by coformulating insulin lispro with treprostinil and ingredients Generally Recognized As Safe (GRAS) by the Food and Drug Administration (FDA) as excipients.

LY900014 is a formulation of insulin lispro that contains the prostacyclin analog treprostinil, citrate, and other excipients. Treprostinil as an excipient enhances the absorption of insulin lispro by local vasodilatation rather than as an active pharmaceutical ingredient that elicits a systemic effect. Treprostinil is a prostacyclin analog administered either by inhalation (Tyvaso®), intravenous (IV) infusion, or continuous SC infusion (Remodulin®) for the treatment of symptomatic pulmonary arterial hypertension, and has been approved in the United States since 2002 (Remodulin package insert, 2014) and in Europe since 2005 (PMR [WWW]). Sodium citrate, an excipient that speeds insulin absorption, is also included in the formulation to further enhance the absorption of insulin lispro. Sodium citrate and the other excipients in the LY900014 formulation are listed in the FDA GRAS food additives database and in the FDA Inactive Ingredients in Approved Drugs database. Furthermore, the excipient concentration in LY900014 is within the limits identified for approved drug products in the FDA Inactive Ingredients in Approved Drugs database.

Please refer to the Humalog local product labeling (for example, Humalog package insert, 2015; Humalog Summary of Product Characteristics, 2016) for more information regarding insulin lispro.

The Investigator's Brochure (IB) describes the clinical and nonclinical development of LY900014.

## 3.3. Benefit/Risk Assessment

More detailed information about the known and expected benefits and risks of insulin lispro may be found in the country-specific product labeling (for example, Patient Information Leaflet, Package Insert, or Summary of Product Characteristics).

Across all doses in the Eli Lilly and Company (Lilly) clinical studies that have evaluated treprostinil as a local vasodilator with or without insulin lispro, there was no clinically significant increase in those adverse events (AEs) associated with systemic absorption of treprostinil, as described in the Remodulin package insert (2014) (that is, headache, diarrhea, nausea, jaw pain, vasodilatation, rash, edema, anorexia, vomiting, asthenia, abdominal pain, and hypotension). The exposures of treprostinil in LY900014 for participants in upcoming and future clinical trials are expected to be much lower than those observed in the dose ranges previously explored with SC bolus administration of treprostinil and are expected to be substantially lower than those observed in the treatment of pulmonary artery hypertension (PAH).

More information about the known and expected benefits, risks, serious AEs (SAEs), and reasonably anticipated AEs of LY900014 can be found in the IB.

# 4. Objectives and Endpoints

Table ITRM.1 shows the objectives and endpoints of the study. Week 52 endpoints for the secondary objectives only apply to the blinded treatment arms of LY900014 and insulin lispro.

Table ITRM.1. Objectives and Endpoints

| | Objectives | | Endpoints |
|---|---|---|---|
| Primar | ry Objective | | - |
| 1. | To test the hypothesis that LY900014 is noninferior to insulin lispro on glycemic control (NIM=0.4% for HbA1c) in patients with T1D, when administered as prandial insulin (0 to 2 minutes prior to the meal), in combination with basal insulin glargine or insulin degludec for 26 weeks | 1. | Difference between LY900014 and insulin lispro in change from baseline to Week 26 in HbA1c |
| Multip | licity Adjusted Objectives | | |
| 2. | To test the hypothesis that LY900014 is superior to insulin lispro in controlling 1-hour PPG excursions, when administered as prandial insulin | 2. | Difference between LY900014 and insulin lispro in the 1-hour PPG excursion (serum glucose measured 1 hour after the start of the meal minus fasting serum glucose) from a MMTT at Week 26 |
| 3. | To test the hypothesis that LY900014 is superior to insulin lispro in controlling 2-hour PPG excursions, when administered as prandial insulin | 3. | Difference between LY900014 and insulin lispro in the 2-hour PPG excursion (serum glucose measured 2 hours after the start of the meal minus fasting serum glucose) from an MMTT at Week 26 |
| 4. | To test the hypothesis that LY900014 is superior to insulin lispro on improving glycemic control (HbA1c) when administered as prandial insulin | 4. | Difference between LY900014 and insulin lispro in change from baseline to Week 26 in HbA1c |
| 5. | To test the hypothesis that LY900014 administered as postprandial insulin 20 minutes after the start of a meal, (LY900014+20), is noninferior to insulin lispro, administered as prandial insulin, on glycemic control (NIM=0.4% for HbA1c) | 5. | Difference between LY900014+20 and insulin lispro in change from baseline to Week 26 in HbA1c |
| Other S | Secondary Objectives | | |
| 6. | To compare LY900014+20 with insulin lispro and LY900014 with respect to 1-hour and 2-hour PPG excursions | 6. | 1- and 2-hour PPG excursions from an MMTT test at Week 26 |
| 7. | To compare the glycemic control of LY900014 with LY900014+20 | 7. | Change from baseline HbA1c values at Week 26 |
| 8. | To compare LY900014, LY900014+20, and insulin lispro on the rate of severe hypoglycemic events | 8. | Rate (events/patient/100 years) of severe<br>hypoglycemic events from baseline through<br>Week 26 and Week 52 |

| Other Secondary Objectives (continued) | |
|---|---|
| 9. To compare LY900014, LY900014+20, and | Rate (events/patient/year and/or |
| insulin lispro with respect to the incidence and | events/patient/30 days) and incidence (percent |
| rate of documented symptomatic postmeal | of patients with at least 1 event) of documented |
| hypoglycemia | symptomatic postmeal hypoglycemia within |
| -31-8-3 | 1 and 2 hours after start of a meal from |
| | Week 12 through Week 26, Week 0 through |
| | Week 26, Week 26 through Week 52, and |
| | Week 0 through Week 52 |
| 10. To compare LY900014, LY900014+20, and | 10. Rate (events/patient/year and/or |
| insulin lispro with respect to the incidence and | events/patient/30 days) and incidence (percent |
| rate of documented symptomatic hypoglycemia | of patients with events) of documented |
| | symptomatic hypoglycemic events from |
| | Week 12 through Week 26, Week 0 through |
| | Week 26, Week 26 through Week 52, and |
| | Week 0 through Week 52 |
| 11. To compare LY900014, LY900014+20, and | 11. Change from baseline 1,5-AG values at |
| insulin lispro with respect to 1,5-AG | Week 26 and Week 52 |
| 12. To compare LY900014, LY900014+20, and | 12. Change from baseline 10-point SMBG values |
| insulin lispro with respect to 10-point SMBG | at Week 26 and Week 52 |
| profiles | at week 20 and week 32 |
| 13. To compare LY900014 , LY900014+20, and | 13. Change from baseline in total, basal and |
| insulin lispro with respect to total, basal, and | prandial insulin doses and prandial/total insulin |
| prandial insulin dose | dose ratios at Week 26 and Week 52 |
| 14. To compare LY900014, LY900014+20, and | 14. Change from baseline in ITSQ regimen |
| insulin lispro with respect to diabetes treatment | inconvenience and lifestyle flexibility domain<br>scores at Week 26 and Week 52 |
| satisfaction as measured by the ITSQ | |
| 15. To compare LY900014, LY900014+20, and | <ol> <li>The proportion of patients with HbA1c &lt;7%<br/>and ≤6.5% at Week 26 and Week 52</li> </ol> |
| insulin lispro with respect to the proportion of | and ≤0.5% at week 20 and week 32 |
| patients achieving HbA1c targets | 16 A-t1 1 C 1 1 t- W1 50 i- |
| 16. To compare the glycemic control of LY900014 | 16. Actual and change from baseline to Week 52 in |
| and insulin lispro | HbA1c |
| Tertiary/Exploratory Objectives | |
| 17. To compare the safety of LY900014, | <ol><li>Adverse events, vital signs, chemistry, and</li></ol> |
| LY900014+20, and insulin lispro | hematology laboratory measures |
| 18. To compare the incidence of treatment- | 18. Incidence of treatment-emergent positive anti- |
| emergent positive anti-insulin lispro antibodies | insulin lispro antibodies |
| for LY900014, LY900014+20, and insulin | • |
| lispro | |
| 21. To compare LY900014, LY900014+20, and | 21. Change in weight (kg) from baseline to |
| insulin lispro with respect to changes in body | Week 26 and Week 52 |
| weight | 11 554 25 445 11 554 52 |
| ··· cagair | 1 |

| Tertiary/Exploratory Objectives (continued) | |
|---|---|
| 22. To compare LY900014, LY900014+20, and | 22. The proportions of patients with shifts in |
| insulin lispro with respect to the proportion of | HbA1c to $<$ 8% and $≤$ 9%, and $>$ 9% from |
| patients achieving improvement from baseline | baseline to Week 26 and Week 52 |
| in HbA1c targets | |
| 23. To compare LY900014, LY900014 +20, and | <ol><li>Within-day and between-day glycemic</li></ol> |
| insulin lispro with respect to glycemic | variability measured by the standard deviation |
| variability | and the coefficient of variation of 10-point |
| | SMBG profiles |

Abbreviations: 1,5-AG = 1,5-Anhydroglucitol; CC

HbA1c = hemoglobin A1c; ITSQ = Insulin Treatment Satisfaction

Questionnaire; MMTT = mixed-meal tolerance test; NIM = noninferiority margin; PPG = postprandial glucose;

SMBG = self-monitored blood glucose; T1D = type 1 diabetes mellitus

# 5. Study Design

# 5.1. Overall Design

Study I8B-MC-ITRM (ITRM) is a Phase 3, prospective, randomized, outpatient, multinational, multicenter, 3-treatment group, parallel, active-controlled study conducted in patients with T1D currently using an MDI regimen. In 2 of the treatment groups, LY900014 and insulin lispro will be administered immediately (0-2 minutes) prior to each meal in a double-blind manner. A third open-label treatment group consists of LY900014 administered 20 minutes after the start of a meal (LY900014+20). It is not possible to blind this treatment group with different injection timing. The study is designed to demonstrate noninferiority of LY900014 when compared with insulin lispro in change from baseline to Week 26 in HbA1c, when both are administered at the start of the meal. For patients in the 2 double-blind arms, the study includes a 1-week screening period and an 8-week lead-in period followed by a 52-week treatment period and a 4-week safety follow-up period. For patients in the open-label treatment group, the treatment period will end after 26 weeks, which will be followed by a 4-week safety follow-up period.

All patients who complete the 4-week safety follow-up visit (Visit 801) and have treatment-emergent insulin lispro antibodies that have not returned to the prespecified baseline range (Visit 2) will be asked to participate in follow-up to monitor insulin lispro antibody levels for up to 26 weeks after Visit 801 as described in Appendix 8.

The purpose of the lead-in period (prior to randomization) will be to titrate basal insulin, obtain preliminary diagnostic laboratory tests, and determine baseline hypoglycemia rates. Patients treated with insulin glargine U-100 (Basaglar/Abasaglar or LANTUS) once or twice daily, insulin glargine U-300 once daily, insulin degludec U-100 or U-200 once daily, insulin detemir U-100 once or twice daily, or neutral protamine Hagedorn (NPH) once or twice daily will be eligible for inclusion in the trial. At Visit 2, patients will be switched to an allowed study basal insulin regimen; insulin glargine U-100 twice daily, insulin glargine U-100 once daily (either in the morning or evening), or insulin degludec U-100 once daily as determined by the investigator. The brand of insulin glargine chosen at Visit 2 should remain the same throughout the study; switching brands should be avoided. Insulin glargine or insulin degludec will be titrated during the 8-week lead-in period using a titration algorithm that should enable patients to reach the target fasting blood glucose (FBG) by the end of this period.

All patients using either insulin aspart or insulin glulisine at screening will be transferred to insulin lispro at Visit 2 so that all patients are using insulin lispro during the lead-in period. Prandial insulin doses or insulin to carbohydrate ratio (ICR), and correction factor (CF) should not be changed during the lead-in period except for safety reasons (hypoglycemia or unacceptable hyperglycemia) or to facilitate basal insulin optimization.

At Visit 8, patients will be randomized to either LY900014 at mealtime, insulin lispro at mealtime, or LY900014 administered 20 minutes after the start of a meal (LY900014+20). During the initial 12 weeks after randomization (intensive titration period), prandial insulin dose should be adjusted as necessary in order to meet the target self-monitored blood glucose (SMBG) levels. Basal insulin may be titrated as needed to facilitate optimal prandial dosing or for safety reasons

such as hypoglycemia or unacceptable hyperglycemia. Thereafter, during the maintenance period (Weeks 12-26 of treatment), it is expected that adjustments to prandial and basal insulin doses would be to maintain glycemic control or for safety reasons such as hypoglycemia or unacceptable hyperglycemia.

For patients continuing into the 26-week long term maintenance period (2 double-blind arms), adjustments to both prandial and basal insulins should be made in order to maintain or further optimize glycemic control, as appropriate.

Figure ITRM.1 illustrates the study design.



Abbreviation: T = telephone visit.

- a At Visit 2, patients on insulin glulisine or insulin aspart will be transferred to insulin lispro. The patients' basal insulin regimen will be switched to insulin glargine U-100 (once or twice daily) or to insulin degludec U-100 once daily. At Visit 8, patients will be randomized to either premeal insulin lispro, premeal LY900014, or LY900014+20 and continue their basal insulin regimen.
- b Titrate basal insulin (see Section 7.2.1.3).
- <sup>c</sup> Titrate prandial insulin (insulin lispro or LY900014) (see Section 7.2.1.4).
- d Patients will discontinue study insulins at Week 26 for the LY900014+20 open-label treatment group or Week 52 for the 2 blinded treatment groups.
- e Eligible patients will have visits at approximately 3-month intervals for up to 26 weeks after Visit 801 for follow-up of insulin lispro antibody levels (see Appendix 8).

Figure ITRM.1. Illustration of study design for Clinical Protocol I8B-MC-ITRM.

## 5.2. Number of Participants

Approximately 1500 participants will be screened to achieve 1199 randomized patients and 1020 patients completing 26 weeks and approximately 646 patients completing 52 weeks (double-blind arms only).

# 5.3. End of Study Definition

End of the study is the last scheduled procedure shown in the Insulin Lispro Antibody Follow-Up Assessment Schedule of Activities (Appendix 8) for the last patient.

# 5.3.1. Safety Follow-Up

Safety follow-up visit guidelines are as follows (see Section 2):

- Patients who discontinue from the study early during the lead-in period (prior to randomization) should complete an early discontinuation visit only.
- Patients who discontinue from investigational product (IP) early but remain in the study should complete all remaining visits per Schedule of Activities, including Visit 801.
- Patients who discontinue from the study early (regardless of whether they discontinue IP at the same time or have discontinued IP at an earlier visit) should complete an early discontinuation visit followed by the safety follow-up visit (Visit 801) per Schedule of Activities.
- Patients in the 2 double-blind arms who finish Visit 22 without early discontinuation of IP should complete a safety follow-up visit (Visit 801) 4 weeks after Visit 22.
- Patients in the open-label treatment group who finish Visit 18 without early discontinuation of IP should complete a safety follow-up visit (Visit 801) 4 weeks after Visit 18.

All patients who complete the 4-week safety follow-up visit (Visit 801) and have treatment-emergent insulin lispro antibodies that have not returned to prespecified baseline range (Visit 2) will be asked to participate in follow-up to monitor insulin lispro antibody levels as described in Appendix 8. Patients participating in the antibody follow-up period will complete the study when insulin antibodies have returned to baseline range or when Visit 803 is completed, whichever occurs first.

# 5.4. Scientific Rationale for Study Design

Study ITRM is a Phase 3 study to evaluate LY900014 compared to insulin lispro each in combination with basal insulin in patients with T1D. The trial has 3 treatment groups, 2 of which are double-blind to allow comparison of LY900014 and insulin lispro when injected at the start of the meal. The third treatment group is open-label due to inability to blind postprandial injection timing of LY900014 (20 minutes after the start of a meal) and will evaluate the efficacy and safety of postprandial dosing. Patients in the 2 blinded arms will continue with double-blind treatment for an additional 26 weeks for a total of 52 weeks to allow comparison of long-term safety and efficacy in a blinded manner. Patients in the open-label treatment group will complete their study participation after the 26-week primary endpoint and safety follow-up.

The study is designed to compare HbA1c lowering as the primary endpoint, a measure of glycemic control accepted by health care providers and regulatory authorities as a validated measure of BG control over time and is the best marker for development and progression of diabetes complications. The lead-in period consists of 8 weeks to allow for optimization of basal insulin dosing. The 26-week treatment period consists of a 12-week intensive titration phase to optimize prandial insulin dosing followed by a 14-week maintenance phase, so the primary endpoint HbA1c reflects glucose control during the 3-month time period when there are minimal changes to insulin dose. The second 26-week period is a long-term maintenance phase to demonstrate durability of glycemic control.

## 5.5. Justification for Dose

LY900014 will have the same insulin lispro concentration (100 U/mL) as that of commercially available Humalog. The addition of treprostinil to the insulin lispro formulation does not modify the physical, chemical, or biological integrity of insulin lispro. The dosage of basal and prandial insulins used in this study should be determined based on the individual needs of each patient.

# 6. Study Population

This study will include patients who have been diagnosed with T1D for at least 1 year, using insulin continuously for at least 1 year, currently on MDI therapy for at least 90 days, and having an HbA1c value of ≥7.0 and ≤9.5% at screening. Patients' basal insulin may be insulin glargine U-100 (Basaglar/Abasaglar or LANTUS) once or twice daily, insulin glargine U-300 once daily, insulin degludec U-100 or U-200 once daily, insulin detemir U-100 once or twice daily, or neutral protamine Hagedorn (NPH) once or twice daily. Patients may be on any approved injectable rapid-acting insulin analog.

Patients must give written informed consent (approved by Lilly or its designee and the ethical review board [ERB] governing the site) before being allowed to participate in the study and before any screening assessments are performed.

Study investigator(s) will review the patient's records and/or history and screening test results/measurements to determine if the patient meets all inclusion and no exclusion criteria to qualify for participation in the study. All screening activities must be completed and reviewed before the patient begins the lead-in period.

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, are not permitted.

## 6.1. Inclusion Criteria

Patients are eligible to be included in the study only if they meet all of the following criteria at screening:

## **Type of Patient and Disease Characteristics**

[1] Men or women diagnosed (clinically) with T1D, based on the World Health Organization (WHO) classification (Appendix 5) for at least 1 year prior to screening, and continuously using insulin for at least 1 year

#### **Patient Characteristics**

- [2] Are at least 18 years of age
- [3] Have been on MDI therapy including a rapid acting insulin analog (insulin lispro U-100, insulin aspart, insulin glulisine) for at least 90 days
- [4] Have been treated for at least 30 days prior to screening with one of the following:
  - a) Insulin glargine U-100 or U-300
  - b) Insulin detemir U-100
  - c) Insulin degludec U-100 or U-200
  - d) NPH
- [5] Have an HbA1c value  $\geq$ 7.0 and  $\leq$ 9.5%, according to the central laboratory at screening (Visit 1).

- [6] Have a body mass index (BMI) of  $\leq$ 35.0 kg/m<sup>2</sup> at screening (Visit 1).
- [7] Male patients:
  - a) No male contraception required except in compliance with specific local government study
- [8] Female patients:
  - a) Women not of childbearing potential may participate and include those who are:
    - i) infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), congenital anomaly such as Mullerian agenesis;

Or

- ii) postmenopausal defined as either
  - (1) a woman 50 to 54 years of age (inclusive) with an intact uterus, not on hormone therapy who has had either
    - (a) cessation of menses for at least 1 year;

Or

(b) at least 6 months of spontaneous amenorrhea with a follicle-stimulating hormone >40 mIU/mL;

Or

(2) a woman 55 or older not on hormone therapy, who has had at least 6 months of spontaneous amenorrhea;

Or

- (3) a woman at least 55 years of age with a diagnosis of menopause prior to starting hormone replacement therapy
- b) Women of childbearing potential participating:
  - i) Cannot be pregnant or intend to become pregnant
  - ii) Cannot be breastfeeding (including the use of a breast pump)
  - iii) Must remain abstinent or use 1 highly effective method of contraception or a combination of 2 effective methods of contraception for the entirety of the study (See Appendix 7)
  - iv) Test negative for pregnancy at the time of screening (Visit 1). Note: a urine pregnancy test is conducted at Visit 8.
- [9] Have access to a telephone or alternative means for close monitoring and communications, and have access to a reliable cellular signal for transmission of the electronic clinical outcomes assessment (eCOA) data

- [10] Have refrigeration in the home or have ready access to refrigeration for storage of insulin therapy
- [11] Patient whom the investigator has determined can be randomized and maintain the treatment regimens based on their previous medical history including insulin dosing regimens, hypoglycemic episodes, and glycemic control
- [12] Capable of, willing, and desirous to do the following:
  - a) Inject insulin with the use of an insulin injection device (insulin pen) according to included directions
  - b) Perform self-BG monitoring including 10-point SMBG on designated days (patients using a personal continuous glucose monitoring [CGM] or flash glucose monitoring [FGM] device for insulin dosing decisions must still use the study glucose meter according to the protocol)
  - c) Keep records in eCOA as required by this protocol
  - d) Participate in two 4-hour mixed-meal tolerance tests (MMTTs) and consume a standardized meal for the tests
  - e) Follow an algorithm for basal insulin adjustment and individualized prandial insulin dosing using fixed pattern adjustment or carbohydrate counting as agreed upon with the investigator
  - f) Comply with the use of the study insulin and scheduled visits
- [13] Considered healthy (apart from T1D) upon completion of medical history, physical examination, vital signs, electrocardiogram (ECG), and analysis of laboratory safety variables, as judged by the investigator

#### **Informed Consent**

[14] Have given written informed consent to participate in this study in accordance with local regulations.

## 6.2. Exclusion Criteria

Patients will be excluded from study enrollment if they meet any of the following criteria at screening:

#### **Medical Conditions**

- [15] Have any other condition (including known drug or alcohol abuse, or psychiatric disorder including eating disorder) that precludes the patient from following and completing the protocol
- [16] Have hypoglycemia unawareness as judged by the investigator
- [17] Have had more than 1 episode of severe hypoglycemia (defined as requiring assistance due to neurologically disabling hypoglycemia) within the last 6 months prior to screening

- [18] Have had more than 1 emergency room visit or hospitalization due to poor glucose control (hyperglycemia or diabetic ketoacidosis) within 6 months prior to screening (Visit 1)
- [19] Have cardiovascular disease within the last 6 months prior to screening, defined as stroke, decompensated heart failure New York Heart Association class III or IV (see Appendix 6), myocardial infarction, unstable angina pectoris, or coronary arterial bypass graft

## [20] Renal:

- a) History of renal transplantation
- b) Currently receiving renal dialysis
- c) Serum creatinine >2.0 mg/dL (177 µmol/L) at screening
- [21] Hepatic: Have obvious clinical signs or symptoms of liver disease (for example, acute or chronic hepatitis, or cirrhosis) or elevated liver enzyme measurements as indicated below at screening (Visit 1):
  - a) Total bilirubin level (TBL)  $\geq$ 2X the upper limit of normal (ULN) (with the exception of Gilberts Disease) as defined by the central laboratory,

OR

b) Alanine aminotransferase (ALT) ≥3X ULN as defined by the central laboratory

OR

- c) Aspartate aminotransferase (AST) ≥3X ULN as defined by the central laboratory
- [22] Malignancy: Have active or untreated malignancy, have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer) for less than 5 years, or are at an increased risk for developing cancer or a recurrence of cancer in the opinion of the investigator
- [23] Have any hypersensitivity or allergy to any of the insulins or excipients used in this trial
- [24] Have hypersensitivity or allergy to any of the ingredients in the standardized test meal (MMTT) (for example, nut allergy)
- [25] Hematologic: Have had a blood transfusion or severe blood loss within 90 days prior to screening or have known hemoglobinopathy, anemia, or any other traits known to interfere with measurement of HbA1c
- [26] Have presence of clinically significant gastrointestinal disease (for example, clinically active gastroparesis associated with wide glucose fluctuations) in the investigator's opinion

[27] Have excessive insulin resistance defined as having received a total daily dose of insulin >1.5 U/kg at the time of screening

## **Prior/Concomitant Therapy**

- [28] Glucocorticoid therapy: Receiving chronic (lasting longer than 14 consecutive days) systemic glucocorticoid therapy (including IV, intramuscular, SC, or oral, but excluding topical, intraocular, intranasal, intra-articular and inhaled preparations) or have received such therapy within 8 weeks immediately prior to screening (Visit 1) with the exception of replacement therapy for adrenal insufficiency
- [29] Have been on a treatment regimen that includes regular human insulin or any premixed insulins within 90 days prior to screening (Visit 1)
- [30] Have used insulin human inhalation powder (Afrezza®) within 90 days prior to screening (Visit 1)
- [31] Have used CSII within the 90 days prior to screening (Visit 1)
- [32] Receiving any oral or injectable medication intended for the treatment of diabetes mellitus other than insulins in the 90 days prior to screening (Visit 1)

## **Prior/Concurrent Clinical Trial Experience**

- [33] Are currently enrolled in any other clinical trial involving an IP or any other type of medical research judged not to be scientifically or medically compatible with this study
- [34] Have participated, within the last 30 days in a clinical trial involving an IP. If the previous IP has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed
- [35] Have previously completed or withdrawn from this study or any other study investigating LY900014 after receiving at least 1 dose of the IP

#### **Other Exclusions**

- [36] Are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
- [37] Are Lilly employees (including employees, temporary contract workers, or designees responsible for the conduct of the study)
- [38] Are unable and/or unwilling to provide informed consent, to make themselves available for the duration of the study, to comply with the use of a data collection device to directly record data, or to abide by study procedures

# 6.3. Lifestyle Restrictions

• Patients should be instructed not to donate blood or blood products during the study.

• Patients should be instructed to avoid major changes in dietary intake or physical activity during the 3 days prior to MMTT.

## 6.4. Screen Failures

Individuals who do not meet the criteria for participation in this study (screen failure) may not be rescreened. Retests are also not allowed, except for cases when results are not available from the original sample.
### 7. Treatments

#### 7.1. Treatments Administered

This study involves a comparison of LY900014 and insulin lispro administered subcutaneously 0 to 2 minutes prior to the start of the meal for 52 weeks. In a third open-label treatment group, LY900014 will be administered postprandially (20 minutes after the start of a meal [LY900014+20]) for 26 weeks. Table ITRM.2 shows the treatment regimens.

Table ITRM.2. Treatment Regimens

| Regimen | Dose<br>Strength | Dose<br>Administration | Route of Administration | Timing of<br>Administration |
|---|---|---|---|---|
| LY900014 | | Individualized<br>dosing | Subcutaneous | 0 to 2 minutes before start of the meal |
| Insulin lispro | | Individualized<br>dosing | Subcutaneous | 0 to 2 minutes before start of the meal |
| LY900014+20 | | Individualized<br>dosing | Subcutaneous | 20 minutes after the start of the meal |

The investigator or his/her designee is responsible for the following:

- explaining the correct use of the IP to the patient including the importance of injection site rotation for both basal and prandial insulin
- explaining requirements for recording insulin doses and injection times to the patient
- verifying that instructions are followed properly
- maintaining accurate records of IP dispensing and collection
- at the end of the study, returning all used and unused IP to Lilly, or its designee, unless the sponsor and sites have agreed all unused medication is to be destroyed by the site, as allowed by local law

# 7.1.1. Packaging and Labeling

Clinical trial materials will be labeled as IP as appropriate, and according to the country's regulatory requirements. Study insulins (LY900014 and insulin lispro) will be supplied by Lilly or its representative, in accordance with current good manufacturing practices, and will be supplied with clinical trial lot numbers. Instruction for Use for the prefilled devices will be provided.

The blinded prefilled pens will contain a concentration of 100 U/mL in 3-mL cartridges of either LY900014 or insulin lispro. The open-label prefilled pens will contain a concentration of 100 U/mL of LY900014.

During the lead-in period, 100 U/mL insulin lispro will be provided using open-label prefilled pens.

#### 7.1.2. Medical Devices

The medical devices provided for use in the study are prefilled pens. LY900014 prefilled pens are new investigational combination products.

## 7.2. Method of Treatment Assignment

Patients who meet all criteria for enrollment will be randomized to double-blind or open-label treatment at Visit 8. Assignment to treatment groups will be determined by a computergenerated random sequence using an interactive web-response system (IWRS). Patients will be randomized to double-blind LY900014, double-blind insulin lispro, or open-label LY900014+20 in a 4:4:3 ratio. Stratification will be by country, HbA1c stratum ( $\leq 7.5\%$ ,  $\geq 7.5\%$  at Visit 7), type of basal insulin during the lead-in period (glargine U-100 or degludec U-100), and prandial insulin dosing plan at randomization (carbohydrate counting, pattern adjustment).

The IWRS will be used to assign all IP during the study, including insulin lispro during the lead-in period. The IWRS will be used to assign prefilled pens containing double-blind IP to each patient randomized to the 2 blinded treatment groups and prefilled pens containing open-label IP to each patient randomized to the LY900014+20 treatment group. Site personnel will confirm that they have located the correct prefilled pens by entering a confirmation number found on the prefilled pens into the IWRS.

# 7.2.1. Selection and Timing of Doses

### 7.2.1.1. Target Glucose Values for Titration of Insulin Therapy

The overall glycemic control goals for all patients enrolled in the study are similar to those recommended by the American Association of Clinical Endocrinologists (AACE) (Bailey et al. 2016). Fasting, prandial, postprandial, and bedtime glucose target values used to reach the SMBG goals and for determination of titration in insulin therapy are listed in Table ITRM.3.

Table ITRM.3. Target Glucose Values for Adjustment of Insulin Therapy

| Time of Target Blood Glucose Measurement | Self-Monitored Blood Glucose (SMBG) Target (Range) |
|---|---|
| Fasting or pre morning meal | Target: 100 mg/dL or 5.6 mmol/L |
| | Range: 80 to <110 mg/dL or 4.4 to 6.1 mmol/L |
| Pre midday meal | Target: 100 mg/dL or 5.6 mmol/L |
| | Range: 80 to <110 mg/dL or 4.4 to 6.1 mmol/L |
| Pre evening meal | Target: 100 mg/dL or 5.6 mmol/L |
| | Range: 80 to <110 mg/dL or 4.4 to 6.1 mmol/L |
| Pre bedtime | Range: 90 to 130 mg/dL or 5.0 to 7.2 mmol/L |
| 1-2 hour postprandial | Target: <140 mg/dL or 7.8 mmol/L |

#### 7.2.1.2. Basal Insulin Therapy

Patients not currently treated with an allowed basal insulin regimen will be transferred at Visit 2 to an allowed study basal insulin regimen (Section 5.1). The initial basal insulin dose may be unit-for-unit of the prestudy basal insulin regimen or 80% of the prior basal insulin daily dose if the patient was previously treated with twice daily NPH or insulin glargine U-300. The basal insulin dose may be influenced by other clinical circumstances and safety considerations known to the investigator; thus, the prescribed basal insulin dose during the study is determined by, and the responsibility of, the investigator. During the study lead-in period, basal insulin doses should be reviewed and adjusted weekly as clinically indicated.

Patients should use the same study basal insulin regimen throughout the trial. The study basal insulin can be dosed at any time during the day and should be taken at approximately the same time of day throughout the course of the study. The patient may be transferred from once daily to twice daily insulin glargine dosing during the lead-in period if needed to reach the FBG target, and should continue the dosing frequency after randomization

#### 7.2.1.3. Basal Insulin Titration

At all clinic and telephone visits during the 8-week lead-in period, basal insulin dose adjustments should be determined by the investigator in discussion with the patient based on SMBG and hypoglycemia data. Additional discussion between visits may be required to enable the patient to reach the FBG target. Patients' basal insulin should be titrated using the titration algorithm to reach the FBG target of 100 mg/dL (5.6 mmol/L). For patients using insulin glargine twice daily, investigators may also consider use of evening premeal SMBG values for assessment of morning insulin glargine dose.

Decreases to the basal insulin dose may be made at any time based upon the judgment of the investigator (for example, in response to hypoglycemia). Modifications in the calculation of the basal insulin dose may also be influenced by other clinical circumstances and safety considerations known to the investigator; thus the prescribed basal insulin dose during the study is determined by, and the responsibility of, the investigator.

Every effort should be made to reach the FBG target during the lead-in period to allow enough time for prandial insulin dose adjustments during the titration period; however, basal insulin dose may be adjusted if needed to facilitate optimal prandial insulin dosing during the intensive titration period (Weeks 0 to 12) or for safety reasons. Thereafter, during the maintenance period (Weeks 12 to 26), it is expected that adjustments to basal insulin doses would be to maintain glycemic control or for safety reasons such as hypoglycemia or unacceptable hyperglycemia. Between Weeks 26 and 52, investigators in discussion with patients should titrate prandial insulin and/or basal insulin as needed in order to maintain or optimize glycemic control.

Assessments of the basal insulin dose should be made at least at weekly intervals based upon the occurrence of hypoglycemia events during the previous week (Table ITRM.4). After the hypoglycemia assessment, the median (or middle) FBG value from the 3 previous corresponding FBG values can be used for basal insulin adjustment as in Table ITRM.5. Additional discussion between visits may be required to enable the patient to reach the FBG target. The basal insulin dose may be adjusted every 3 to 4 days (twice per week) when appropriate, based on the

patient's glycemic needs and SMBG levels. Investigators may use discretion and provide direction for patients to adjust the basal insulin dose. For patients treated with twice daily insulin glargine, the evening premeal SMBG level may be evaluated for assessment of the morning dose of insulin glargine.

Table ITRM.4. Basal Insulin Hypoglycemia Assessment

| Hypoglycemic Events in the Previous Week | Basal Insulin Change (units) |
|---|---|
| 2 or more nocturnal hypoglycemia events occur or 1 severe | Titrate the basal dose down to the previous basal |
| hypoglycemia event occurs at any time of the day | insulin dose (or by 10% if this is first dose) |
| 1 maghine al himaghia and a come | Do not increase basal insulin dose and consider |
| 1 nocturnal hypoglycemia event occurs | reducing the dose if clinically indicated |
| | Titrate the basal insulin up based upon the median |
| No nocturnal events occur | FBG for the previous 3 FBG values. See |
| | Table ITRM.5 |

Abbreviation: FBG = fasting blood glucose.

Table ITRM.5. Summary of Basal Insulin Adjustments after Hypoglycemia Assessment

| | When Basal Insulin ≤14 units | When Basal Insulin ≥15 units |
|---|---|---|
| If median (middle) FBG | Adjust the basal dose by: | Adjust the basal dose by: |
| from the 3 previous FBG | | |
| values is: | | |
| ≤70 mg/dL | Decreasing dose to previous lower dose <sup>a</sup> | Decreasing dose to previous lower dose <sup>a</sup> |
| (≤3.9 mmol/L) | | |
| 71–100 mg/dL | No adjustment | No adjustment |
| (>3.9–5.6 mmol/L) | | |
| 101–139 mg/dL | Increasing by 1 unit | Increasing by 2 units |
| (>5.6–7.7 mmol/L) | | |
| 140–179 mg/dL | Increasing by 2 units | Increasing by 3 units |
| (>7.8–9.9 mmol/L) | | |
| ≥180 mg/dL | Increasing by 3 units | Increasing by 4 units |
| (≥10 mmol/L) | | |

Abbreviation: FBG = fasting blood glucose.

Source: Adapted from Bartley et al. 2008 and Bolli et al. 2009.

#### 7.2.1.4. Study Prandial Insulin Therapy

Patients treated with insulin aspart or insulin glulisine as their prestudy prandial insulin will be transferred to insulin lispro (unit for unit) at Visit 2. Insulin lispro will be dispensed to all patients for use throughout the lead-in period.

Patients will be randomized (Visit 8) to either LY900014 at mealtime, insulin lispro at mealtime, or LY900014 administered 20 minutes after the start of a meal (LY900014+20). Patients will administer their first study prandial insulin with the next meal following the baseline MMTT.

<sup>&</sup>lt;sup>a</sup> If there is no previous dose because this was the first assigned dose after randomization, then the basal dose should be decreased by 10% in consultation with the investigator.

Patients should have 3 doses of prandial insulin per day and eat 3 main meals per day (morning, midday, and evening) on a regular basis. Patients may also eat a snack and cover with bolus insulin if that is their usual practice.

This study will use 2 possible plans for determining prandial insulin dosing including:

- Pattern adjustment: The patient is prescribed a fixed dose or dose range of insulin for each meal. The fixed insulin dose may be individualized for each meal.
- Carbohydrate counting: The patient performs carbohydrate counting for prandial insulin dosing (ICR plan) and prandial insulin dose is based upon the estimated carbohydrate content of the meal (as unit insulin per grams carbohydrate).

Carbohydrate counting is the preferred method for determining prandial insulin dosing requirements. For patients entering the study using the pattern adjustment method, education and training may be provided at the start of and throughout the 8-week lead-in period to teach willing and desirous patients how to effectively use the carbohydrate counting method for determining meal time insulin doses. Patients who have demonstrated proficiency with carbohydrate counting in the opinion of the investigator should continue using this method during the treatment period.

The patient should maintain the same prandial insulin dosing plan throughout the study. In order to account for potential differences between patients who manage prandial insulin doses using pattern adjustment and those who use carbohydrate counting, stratification by patients' prandial insulin dosing plan will ensure balance of this factor across treatments. Correction factor(s) (for example, 1 unit of insulin per glucose [mg/dL or mmol/L] above target goal) may be implemented with either prandial insulin dosing plan. Adjustments in insulin dosage should also take into account conditions of stress and/or exercise and should be made individually.

At randomization (Visit 8), the starting study insulin doses may be initiated unit for unit; however, investigators may consider reducing the prandial or correction insulin doses by approximately 10 to 20% based on the patient's overall glycemic status or other considerations known to the investigator in order to reduce the risk of postprandial hypoglycemia.

For patients who are <u>carbohydrate counting</u>, the insulin to carbohydrate ratio and correction factor should be assessed and adjusted as needed, at least weekly, in order to meet the target SMBG levels described in Table ITRM.5 during the initial 12 weeks after randomization (the intensive titration period). The insulin to carbohydrate ratio may be adjusted every 3 to 4 days (twice per week) when appropriate, based on the patient's glycemic needs and SMBG levels. Postprandial SMBG levels from 10-point SMBG profiles should also be evaluated for optimization of prandial insulin dosing.

Additional 2-hour postprandial SMBG monitoring should be considered during the days following transition to study insulin beginning at Visit 8. During the maintenance period, Weeks 12 to 26 it is expected that prandial insulin dose adjustments would be to maintain glycemic control or for safety reasons such as hypoglycemia or unacceptable hyperglycemia; however, if SMBG targets have not been achieved, titration of prandial insulin should continue. Between

Weeks 26 and 52, investigators in discussion with patients should titrate prandial insulin as needed in order to maintain or optimize glycemic control.

For patients who are using pattern adjustment, the prandial insulin dose should be assessed and adjusted as needed 1 to 2 times each week, and the correction factor should be assessed and adjusted weekly as needed during the initial 12 weeks after randomization (the intensive titration period). In addition to the weekly investigator dose assessment, investigators may use discretion and encourage patients to make 1 additional prandial insulin dose adjustments for a maximum of 2 prandial adjustments per week. During the maintenance period (Weeks 12-26), prandial insulin dose adjustments should be made in order to maintain glycemic control and for safety reasons such as hypoglycemia or unacceptable hyperglycemia; however, if glycemic and SMBG targets have not been achieved, titration of prandial insulin should continue. Between Weeks 26 and 52, investigators in discussion with patients should titrate prandial insulin as needed in order to maintain or optimize glycemic control. Modifications in the calculation of the insulin dose may also be influenced by other clinical circumstances and safety considerations known to the investigator. Therefore, the prescribed prandial insulin dose is determined by, and the responsibility of, the investigator.

In the pattern adjustment plan, assessment of the prandial insulin dose includes review of the previous 3 to 7 days of SMBG levels for the corresponding meal or bedtime (Table ITRM.6). For example, if assessing the need to adjust the fasting (pre morning meal) prandial insulin dose, review the preceding 3 to 7 pre midday meal SMBG levels.

Table ITRM.6. Prandial Insulin Doses and Corresponding Self Monitored Blood Glucose Values Pattern Adjustment Plan

| Prandial Insulin Dose Assessed | Corresponding SMBG Values for Review |
|--------------------------------|------------------------------------------|
| Fasting or morning premeal | 3-7 previous midday premeal SMBG values |
| Midday premeal | 3-7 previous evening premeal SMBG values |
| Evening premeal | 3-7 previous bedtime SMBG values |

Abbreviation: SMBG = self-monitored blood glucose.

The median (or middle) value from premeal glucose readings from the 3 to 7 previous days is chosen as the "adjustment value" and the change in dose (either increase or decrease) is based upon this value (Table ITRM.7).

| Table ITRM.7. | LY900014 or Insulin Lispro Adjustment Algorithm Pattern |
|---------------|---------------------------------------------------------|
| | Adjustment Plan |

| If Meal Time Dose of | Median SMBG Value | Median SMBG Value at | Median SMBG Value |
|---|---|---|---|
| Insulin Lispro is: | Below Target Range | Target Rangea | Above Target Range |
| <u>≤</u> 10 units | Decrease by 1 unit | No change | Increase by 1 unit |
| 11–19 units | Decrease by 2 units | No change | Increase by 2 units |
| ≥20 units | Decrease by 3 units | No change | Increase by 3 units |

Abbreviation: SMBG = self-monitored blood glucose.

a Median SMBG value at target range OR experienced 1 unexplained hypoglycemic event (≤70 mg/dL

[3.9 mmol/L] or signs/symptoms consistent with hypoglycemia noted.

Target Range: Premeal: 80-130 mg/dL or 4.4-7.2 mmol/L Bedtime: 90-130 mg/dL or 5.0-7.2 mmol/L.

Source: Adapted from Bergenstal et al. 2008.

Patients who wear their personal CGM/FGM device prior to study entry will be allowed to continue to wear their CGM/FGM device during the study. However, these patients should be instructed to perform SMBG monitoring using the study glucose meter according to the protocol. Investigators must use the SMBG levels to make treatment decisions.

#### 7.2.1.5. Transitioning off Study Prandial Insulin Therapy

Patients in the 2 blinded arms should take their last dose of study insulin (LY900014 or insulin lispro) at Visit 22 or at early discontinuation.

Patients in the open-label treatment group, LY900014+20, should take their last dose of study insulin at Visit 18 with the MMTT or at early discontinuation.

No special instructions for transition to nonstudy prandial insulin are necessary for patients who were randomized to either LY900014 or insulin lispro. After completion of study treatment patients will restart the prandial insulin therapy used prior to study entry. Additional guidance for insulin therapy after the treatment period is provided in Section 7.8.2 and Appendix 8.

# 7.3. Blinding

This is a double-blind study in which 2 of the treatment arms, LY900014 and insulin lispro, will be administered immediately (0-2 minutes) prior to each meal in a double-blind manner. Investigators, patients, and study site personnel will be blinded to assigned dosing regimens throughout the study. A third open-label treatment group consists of LY900014 administered 20 minutes after the start of a meal (LY900014+20)

To preserve the blinding of the study, the Lilly study team will be blinded to double-blind treatment assignments until after the primary endpoint database lock. A limited number of study team members will have access to the unblinded treatment assignments and unblinded data at the time of the primary endpoint database lock. The primary endpoint database lock is planned to occur after all patients in the double-blind treatment groups have completed or discontinued the study prior to Visit 18 and after all patients in the open-label treatment group have completed Visit 801. Investigators, site staff, clinical monitors, patients, and study team members who

interact directly with site personnel after primary endpoint database lock will remain blinded to the treatment assignments until the study is complete.

Emergency unblinding for AEs may be performed through the IWRS, which may supplement or take the place of emergency codes generated by a computer drug-labeling system. This option may be used ONLY if the patient's well-being requires knowledge of the patient's treatment assignment. Unblinding events are recorded and reported by the IWRS.

If an investigator, site personnel performing assessments, or patient is unblinded, the patient must be discontinued from IP and should remain in the study.

In case of an emergency, the investigator has the sole responsibility for determining if unblinding of a patient's treatment assignment is warranted. Patient safety must always be the first consideration in making such a determination. If the investigator decides that unblinding is warranted, the investigator should make every effort to contact the Lilly clinical research physician (CRP/CRS) prior to unblinding a patient's treatment assignment unless this could delay emergency treatment of the patient. If a patient's treatment assignment is unblinded, Lilly must be notified immediately.

# 7.4. Dosage Modification

See Section 7.2.1.

# 7.5. Preparation/Handling/Storage/Accountability

The investigator or his/her designee is responsible for confirming appropriate temperature conditions have been maintained during transit for all study treatment received and any discrepancies are reported and resolved before use of the study treatment.

Only patients enrolled in the study may receive IP, and only authorized site staff may supply or administer study treatment. All study treatments should be stored in an environmentally controlled and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the investigator and authorized site staff.

All insulin products must be stored at the investigative site under refrigerated conditions (between 2°C and 8°C) in a locked and secure place. Insulin must not be frozen.

In-use insulins should be maintained at room temperature, and refrigerated material should be warmed to near room temperature before injection. In-use insulin must not be used after 28 days.

The investigator is responsible for study treatment accountability, reconciliation, and record maintenance (such as receipt, reconciliation, and final disposition records).

# 7.6. Treatment Compliance

The investigator or designee will assess compliance of the patient at each visit, based on a review of the patient's glycemic control, adherence to the visit and treatment schedule, and completion of patient eCOA. Patients who are deemed noncompliant will receive additional diabetes

education and training, as required, and the importance of compliance with the protocol will be reinforced. Patients who, in the opinion of the investigator, are deemed consistently noncompliant may be discontinued from IP or from the study. The prandial insulin dose times and meal times will be collected for assessing compliance of the timing of prandial insulin administration relative to meal time (premeal and postmeal).

### 7.7. Concomitant Therapy

Guidance on restrictions for concomitant therapies is provided in Table ITRM.8.

Table ITRM.8. Concomitant Medications

| Drug Class | Acute<br>Use | Chronic<br>Use | Safety Follow-Up and<br>Insulin Lispro Antibody | Conditions |
|---|---|---|---|---|
| NPH, insulin glargine U-300, insulin detemir, insulin degludec U-200 | No | No | Yes | |
| Regular human insulin | No | No | No | |
| Afrezza® (inhaled insulin), or premixed human or premixed analog insulin | No | No | No | |
| Any noninsulin diabetes treatment therapy | No | No | No | |
| Systemic glucocorticosteroid (including IV, intramuscular, SC, or oral but excluding topical, inhaled, intraocular, intra-articular, or intranasal preparations) | Yes | No | No | During the lead-in period, allow 1-time use for ≤7 consecutive days. During all other study periods, allow 1-time use for ≤14 consecutive days. |

Abbreviations: IV = intravenous; NPH = neutral protamine Hagedorn; SC = subcutaneous.

# 7.8. Treatment after the End of the Study

#### 7.8.1. Continued Access

LY900014 will not be made available to patients after conclusion of the study. Rapid-acting insulin analogs are available in all countries for use as prandial insulin.

# 7.8.2. Special Treatment Considerations

After discontinuation of IP at the end of the treatment period or earlier, randomized patients should restart the prandial insulin used prior to study entry. Patients may remain on the basal insulin used during the study (if it was changed at Visit 2) at the discretion of the investigator or return to their prestudy basal insulin. Please also refer to Appendix 8 for information regarding the insulin lispro antibody follow-up assessment.

Investigators should provide patients with appropriate guidance for glucose monitoring and insulin dose adjustment throughout the follow-up period in order to maintain glycemic control.

### 8. Discontinuation Criteria

## 8.1. Discontinuation from Study Treatment

In the event that a patient is discontinued from the study treatment, the investigator should encourage the patient to remain in the study for continued safety monitoring.

Lilly recognizes the importance of complete data collection. This study includes elements to minimize missing data. Randomized patients who are discontinued from IP before study completion are encouraged to remain in the study for continued monitoring. For patients who remain in the study after early discontinuation of IP, both efficacy (including HbA1c) and safety data will be collected at scheduled visits. The difference between stopping IP and discontinuing the study will be explained to patients as part of the informed consent, and patients will be encouraged to continue in the study even if they stop study drug. In addition, study site investigators will be trained on the importance of complete data collection, with additional reeducation of sites and patients as necessary.

### 8.1.1. Permanent Discontinuation from Study Treatment

Patients will be discontinued from the IP in the following circumstances:

- The investigator may decide that the patient should stop IP. If this decision is made because of an AE, SAE, or a clinically significant laboratory value, the study drug is discontinued for that patient and appropriate measures are to be taken. Lilly or its designee is to be alerted.
- The patient may decide to stop IP.
- If the patient becomes pregnant.
- If an investigator, study site personnel performing assessments, or patient is unblinded, the patient must discontinue IP.
- If the patient, for any reason, requires treatment with another therapeutic regimen or therapeutic agent that has been demonstrated to be effective for treatment of the study indication. Discontinuation from IP should occur prior to introduction of the new agent.
- Use of prohibited concomitant medication, see Table ITRM.8.
- Patient has not taken IP for more than 14 consecutive days.

Discontinuation of the IP for abnormal liver tests **should be considered** by the investigator when a patient meets one of the following conditions after consultation with the Lilly designated medical monitor:

- ALT or AST >8X ULN.
- ALT or AST >5X ULN for more than 2 weeks.
- ALT or AST >3X ULN and total bilirubin level(TBL) >2X ULN or prothrombin time >1.5X ULN.

- ALT or AST >3X ULN with the appearance of fatigue, nausea, vomiting, right upper-quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%).
- alkaline phosphatase (ALP) >3X ULN.
- ALP >2.5X ULN and TBL >2X ULN.
- ALP >2.5 ULN with the appearance of fatigue, nausea, vomiting, right upper-quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%).

## 8.1.2. Temporary Discontinuation from Study Treatment

During the study, patients who temporarily discontinue the IP may be able to resume IP based on the following scenario.

Patient has not taken IP for 14 consecutive days or less:

• If the treatment regimen restarts within 14 days of when the patient initially stopped taking IP, patient may continue in the study and begin treatment again with IP. During this time, nonstudy insulins may have been used. If the patient decides to continue in the study, no early termination procedures will be completed. Patients will continue study visits through the safety follow-up.

## 8.1.3. Discontinuation of Inadvertently Enrolled Patients

If the sponsor or investigator identifies a patient who did not meet enrollment criteria and was inadvertently enrolled, a discussion must occur between the sponsor CRP and the investigator to determine if the patient may continue in the study. If both agree it is medically appropriate to continue, the investigator must obtain documented approval from the sponsor CRP to allow the inadvertently enrolled patient to continue in the study with or without treatment with IP.

# 8.2. Discontinuation from the Study

Some possible reasons that may lead to permanent discontinuation include:

- Enrollment in any other clinical trial involving an IP or enrollment in any other type of medical research judged not to be scientifically or medically compatible with this study
- Participation in the study needs to be stopped for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and good clinical practice (GCP)
- The investigator decides to discontinue the patient from the study
- The patient requests to be discontinued from the study
- The patient discontinues insulin lispro or study-allowed basal insulin regimen for >14 consecutive days in the lead-in period.

Patients who discontinue the study early, but after randomization, will have early discontinuation procedures performed as shown in the Schedule of Activities (Section 2).

Patients who discontinue during the lead-in period will not need to fast, have laboratory tests drawn, or complete questionnaires, but will have all other early discontinuation procedures performed.

## 8.3. Lost to Follow-Up

A patient will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site. Site personnel are expected to make diligent attempts to contact patients who fail to return for a scheduled visit or were otherwise unable to be followed up by the site.

# 9. Study Assessments and Procedures

Section 2 lists the Schedule of Activities, with the study procedures and their timing (including tolerance limits for timing).

Appendix 2 lists the laboratory tests that will be performed for this study.

Unless otherwise stated in the subsections below, all samples collected for specified laboratory tests will be destroyed within 60 days of receipt of confirmed test results. Certain samples may be retained for a longer period, if necessary, to comply with applicable laws, regulations, or laboratory certification standards.

### 9.1. Efficacy Assessments

## 9.1.1. Primary Efficacy Assessments

The primary efficacy measure is the change from baseline to Week 26 in HbA1c.

## 9.1.2. Secondary Efficacy Assessments

The following secondary efficacy measures will be collected at the times shown in the Schedule of Activities (Section 2).

- Fasting and PPG collected during the MMTT
  - o 1-hour and 2-hour PPG excursions: serum glucose measured 1 hour and 2 hours after the start of a meal minus fasting serum glucose
  - o Incremental areas under the serum glucose concentration-time curve from 0 to 30 minutes, 0 to 1 hour, 0 to 2 hours, 0 to 3 hours, and 0 to 4 hours after a meal; maximum serum glucose after a meal
  - Glucose variability measured by the coefficient of variation and standard deviation (SD)
- 1,5-Anhydroglucitol (1,5-AG)
- SMBG 10-point profiles (fasting, 1 hour post morning meal, 2 hours post morning meal, pre midday meal, 1 hour post midday meal, 2 hours post midday meal, pre evening meal, 1 hour post evening meal, 2 hours post evening meal, and bedtime)
  - 1-hour and 2-hour PPG excursions
  - Within- and between-day glucose variability measured by the coefficient of variation and SD
- Proportion of patients with HbA1c  $\leq$ 6.5% and  $\leq$ 7.0%
- Prandial, basal, and total insulin dose (units and units/kg), and prandial/total insulin ratio

### 9.1.3. Appropriateness of Assessments

All efficacy and safety assessments included in this study are generally regarded as reliable and accurate with respect to diabetes mellitus.

## 9.1.4. Study Procedures

The following procedures will be performed at the times shown in the Schedule of Activities (Section 2).

#### 9.1.4.1. Electronic Clinical Outcomes Assessment

The eCOA diary will wirelessly receive all glucose data directly from the BG meters, thereby increasing the validity of measures reported by the patient and minimizing transcription errors in recording the measures. The use of e-diaries should also allow more complete and accurate capturing of hypoglycemia events, as well as more frequent and timely interactions between investigator and patients as the intensity of their individual diabetes management increases.

The system will be used to collect time of the meal and prandial insulin doses (date, time, and actual dose taken) and the basal insulin dose, 3 days prior to study visits, on the days of 10-point SMBG profiles and at other times as clinically indicated. For patients who are carbohydrate counting, the grams of carbohydrate will be entered for each meal during the 10-point SMBG profile days. Hypoglycemic events will be captured throughout the clinical study in eCOA along with date and time of the BG level if measured and hypoglycemia treatment and outcome data. Additionally, the eCOA system will incorporate study-specific reminders for patients to perform the 10-point SMBG profiles.

Physicians and designated clinical staff will have access via eCOA portal (secure web-based site), to the ongoing near real-time updating of the BG readings, insulin doses administered, hypoglycemic events, and dosing time relative to the meal. Manual inspection of data will support at least weekly patient monitoring as an enhancement to standard of care for patient safety, as well as the potential for reaching an optimum efficacy outcome. Investigative staff will assess clinical data via the eCOA portal and recommend adjustments in basal and prandial insulin (also refer to Section 7.2.1).

An instruction manual will be provided to patients and investigative sites. Additional instruction and training will be provided to the investigative sites regarding data collection, review, retention and archival processes. In the event of eCOA e-diary malfunction or loss, the patient will be instructed to immediately contact the investigative site for instructions regarding replacement of the equipment.

#### 9.1.4.2. Four-Point Self-Monitoring Blood Glucose

Patients should be instructed to measure a minimum of 4 SMBG readings daily (consists of fasting [pre morning meal], pre midday meal, pre evening meal, and pre bedtime), with additional readings as needed for glucose self-management. Site personnel may request additional BG monitoring from patients and/or assess BG values at other times (such as postprandial BG measurements) to make clinical management decisions. Missing values in 4-

point SMBG profiles will not be considered protocol deviations unless, in the opinion of the investigator, they are excessive and reflect noncompliance with the protocol.

### 9.1.4.3. Ten-Point Self-Monitoring Blood Glucose

Patients in all 3 study arms should be instructed to perform 10-point SMBG profiles prior to 5 visits during the study (Visits 8, 11, 13, 15, and 18). Patients in the 2 blinded arms will perform 10-point SMBG profiles prior to 2 additional visits, Visits 20 and 22. Three 10-point profiles should be done during the 2 weeks prior to each visit. Each 10-point profile during this 2-week time interval should be completed over a 1-day period, preferably on 3 nonconsecutive days (weekdays and weekends) per Section 2. The 10-point profile consists of 10 SMBG measurements on the same day at premeal; 1 hour and 2 hours after the start of the morning, midday, and evening meals; and at bedtime. The 10-point SMBG profile is inclusive of the daily 4-point SMBG readings. Patients should be encouraged to eat a morning, midday, and evening meal on the days that the 10-point SMBG is monitored. Premeal measurements should be taken before the patient begins eating the meal. Patients may eat a snack and cover with bolus insulin if that is their usual practice. Missing values in 10-point SMBG profiles will not be considered protocol deviations unless, in the opinion of the investigator, they are excessive and reflect noncompliance with the protocol.

#### 9.1.4.4. Mixed-Meal Tolerance Test

A 4-hour MMTT will be performed in all patients at baseline (Week 0, Visit 8) and at the end of the 26 weeks of treatment (Visit 18). Patients will be instructed to fast for at least 8 hours prior to the administration of the MMTT at the study site.

The MMTT can occur 0 to 4 days prior to the visit. The MMTT can be rescheduled up to 2 times within the visit window, ideally at 24-hour intervals, if the patient does not meet the target FBG. It is preferred for the rescheduled MMTT to occur as close to the visit date as possible.

**Target FBG prior to the MMTT**: Patients must have an FBG in the range of 71 to 180 mg/dL (3.9-10.0 mmol/L) prior to starting the MMTT. If the glucose is outside of this range, the MMTT should be rescheduled

In order to increase the likelihood of having patients arrive on the morning of the MMTT within the target FBG range, please note the following:

- Patients should be instructed to avoid major changes in dietary intake or physical activity during the 3 days prior to the MMTT.
- Patients should be instructed to inject basal insulin according to their usual schedule.
- Patients should not administer correction doses with insulin lispro or LY900014 within 4 hours of the start of the MMTT.

During the 8-hour fasting period and up to 2 hours prior to the start of the MMTT, episodes of non-severe hypoglycemia (symptoms or BG  $\leq$ 70 mg/dL [3.9 mmol/L]) can be treated with 15 to 20 grams of carbohydrate. If a hypoglycemic episode requires more than approximately 20 grams of carbohydrate within 8 hours of the start of the MMTT or the patient experiences a

severe hypoglycemic episode (as defined in Sections 9.4.1 and 9.4.2), the patient should be instructed to notify the site and the MMTT must be rescheduled.

**Test Meal**: The MMTT meal (approximately 700 kcal and 100 grams of carbohydrate) will consist of a liquid nutrition shake(s) (such as Ensure Plus®, Abbott Nutrition). Patients are expected to consume the meal within 15 minutes. Patients should consume the same test meal for both the baseline and end of primary treatment period MMTT, if possible.

**Insulin Injection**: During the Visit 8 MMTT, all patients will have insulin lispro injected 0 to 2 minutes before the start of the meal. During the Visit 18 MMTT, patients randomized to either of the 2 blinded arms will have their blinded study insulin, either LY900014 or insulin lispro, injected 0 to 2 minutes before the start of the meal. Patients randomized to the LY900014+20 treatment group will have LY900014 injected at 20 minutes after the start of the MMTT. The prandial insulin dose administered during the MMTT will be individualized for each patient.

- If the patient uses the carbohydrate counting prandial dosing plan, the morning meal ICR will be used to calculate the prandial insulin dose for the MMTT.
- If the patient does not use carbohydrate counting, the prandial insulin dose for the MMTT should be calculated based on the average total daily insulin dose for the 3 days prior to the MMTT per Table ITRM.9.
- Modifications in the calculation of the insulin dose may also be influenced by other clinical circumstances and safety considerations known to the investigator; thus the MMTT prandial insulin dose is determined by, and the responsibility of, the investigator.

Table ITRM.9. Insulin to Carbohydrate Ratio for Determining the Prandial Insulin dose for the Mixed-Meal Tolerance Test: For Use with Patients who use Pattern Adjustment to Determine Prandial Insulin Doses

| Average Total (Basal+Bolus) Insulin Dose | Insulin to Carbohydrate Ratio |
|---|---|
| (units) in the Last 3 Days | (1 unit per number of grams carbohydrate) |
| 8-11 units | 1 unit : 50 grams |
| 12-14 | 1:40 |
| 15-18 | 1:30 |
| 19-21 | 1:25 |
| 22-27 | 1:20 |
| 28-35 | 1:15 |
| 36-45 | 1:12 |
| 46-55 | 1:10 |
| 56-65 | 1:8 |
| 66-80 | 1:6 |
| 81-120 | 1:5 |
| >120 | 1:4 |

Source: Scheiner [WWW].

**Hypoglycemia during the MMTT**: If a patient has signs or symptoms of hypoglycemia during the MMTT, BG should be measured with a glucometer. If the patient's BG is  $\leq$ 70 mg/dL (3.9 mmol/L), then the patient should receive 15 grams of rapidly absorbable oral carbohydrate. The patient's BG should be retested in 15 minutes or as clinically indicated, and if still  $\leq$ 70 mg/dL (3.9 mmol/L), treatment with another 15 grams of carbohydrate should be given until BG is  $\geq$ 70 mg/dL (3.9 mmol/L). Sample collection should continue per the schedule if possible.

**Sample Collection**: Time 0 of the MMTT will be when the patient starts to consume the meal. Serial venous blood samples to measure serum glucose will be taken at time -15, 0, 15, 30, 60, 120, 180, and 240 minutes after the start of the meal.

#### 9.1.4.5. Diabetes Education and Nutritional Counseling

Initial training at Visit 2 will include diabetes education and nutrition counseling as well as hypoglycemia recognition and management. Appropriate site personnel will administer training and education using locally approved diabetes education/training materials and programs or by using other materials that may be provided by the sponsor. Patients may be provided abbreviated training and education at visits following Visit 2 based upon patient needs.

#### 9.2. Adverse Events

Investigators are responsible for monitoring the safety of patients who have entered this study and for alerting Lilly or its designee to any event that seems unusual, even if this event may be considered an unanticipated benefit to the patient.

The investigator is responsible for the appropriate medical care of patients during the study.

Investigators must document their review of each laboratory safety report.

The investigator remains responsible for following, through an appropriate health care option, AEs that are serious or otherwise medically important, considered related to the IP or the study, or that caused the patient to discontinue the IP before completing the study. The patient should be followed until the event resolves, stabilizes with appropriate diagnostic evaluation, or is reasonably explained. The frequency of follow-up evaluations of the AE is left to the discretion of the investigator.

Lack of drug effect is not an AE in clinical studies, because the purpose of the clinical study is to establish treatment effect.

After the informed consent form (ICF) is signed, study site personnel will record via electronic data entry the occurrence and nature of each patient's preexisting conditions, including clinically significant signs and symptoms of the disease under treatment in the study. In addition, site personnel will record any change in the condition(s) and any new conditions as AEs. Investigators should record their assessment of the potential relatedness of each AE to protocol procedure and/or IP, via electronic data entry.

The investigator will interpret and document whether or not an AE has a reasonable possibility of being related to study treatment, study device, or a study procedure, taking into account the disease, concomitant treatment, or pathologies.

A "reasonable possibility" means that there is a cause and effect relationship between the IP, study device, and/or study procedure and the AE.

The investigator answers yes/no when making this assessment.

Planned surgeries and nonsurgical interventions should not be reported as AEs unless the underlying medical condition has worsened during the course of the study.

If a patient's IP is discontinued as a result of an AE, study site personnel must report this to Lilly or its designee via electronic data entry, clarifying if possible, the circumstances leading to any dosage modifications or discontinuations of treatment.

#### 9.2.1. Serious Adverse Events

An SAE is any AE from this study that results in one of the following outcomes:

- Death
- Initial or prolonged inpatient hospitalization
- A life-threatening experience (that is, immediate risk of dying)
- Persistent or significant disability/incapacity
- Congenital anomaly/birth defect
- Considered significant by the investigator for any other reason: important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious, based upon appropriate medical judgment.
- When a condition related to the prefilled pen necessitates medical or surgical intervention to preclude either permanent impairment of a body function or permanent damage to a body structure, the serious outcome of "required intervention" will be assigned.
- Severe hypoglycemia events: episodes of severe hypoglycemia as determined by the investigator according to the definition provided in Sections 9.4.1 and 9.4.2 must be reported as SAEs.

Although all AEs occurring after signing the ICF are recorded in the case report form (CRF), SAE reporting begins after the patient has signed the ICF and has received IP. However, if an SAE occurs after signing the ICF, but prior to receiving IP, it needs to be reported ONLY if it is considered reasonably possibly related to study procedure.

Study site personnel must alert Lilly or its designee of any SAE within 24 hours of investigator awareness of the event via a sponsor-approved method. If alerts are issued via telephone, they are to be immediately followed with official notification on study-specific SAE forms. This 24-hour notification requirement refers to the initial SAE information and all follow-up SAE information.

Pregnancy (during maternal or paternal exposure to IP) does not meet the definition of an AE. However, to fulfill regulatory requirements, any pregnancy should be reported following the SAE process to collect data on the outcome for both mother and fetus.

Investigators are not obligated to actively seek AEs or SAEs in patients once they have discontinued and/or completed the study (the patient summary CRF has been completed). However, if the investigator learns of any SAE, including a death, at any time after a patient has been discharged from the study, and the investigator considers the event reasonably possibly related to the study treatment or study participation, he/she must promptly notify Lilly.

#### 9.2.1.1. Suspected Unexpected Serious Adverse Reactions

Suspected unexpected serious adverse reactions (SUSARs) are serious events that are not listed in the IB and that the investigator identifies as related to IP or procedure. United States 21 CFR 312.32 and European Union Clinical Trial Directive 2001/20/EC and the associated detailed guidance or national regulatory requirements in participating countries require the reporting of SUSARs. Lilly has procedures that will be followed for the recording and expedited reporting of SUSARs that are consistent with global regulations and the associated detailed guidance.

## 9.2.2. Complaint Handling

Lilly collects product complaints on IPs and drug delivery systems used in clinical studies in order to ensure the safety of study participants, monitor quality, and to facilitate process and product improvements.

Patients will be instructed to contact the investigator as soon as possible if he or she has a complaint or problem with the IP and/or drug delivery system so that the situation can be assessed.

- Complaints must be reported by site staff <u>within 24 hours</u> of notification to the clinical site/study personnel, or <u>within 24 hours</u> of study/site personnel becoming aware of a product issue, regardless of the availability of the complaint sample.
- Retain the IP under appropriate storage conditions, if available or when obtained, until instructed to return it to Lilly.
- Product complaints for non-Lilly Products (including concomitant drugs) that do not have a Lilly Product Batch or Control number, are reported <u>directly to the manufacturer per product label</u>.
- Follow the instructions outlined in the Product Complaint Form for other reporting requirements.

#### 9.3. Treatment of Overdose

Excess insulin administration may result in hypoglycemia. Refer to the IB for LY900014 and product label for insulin lispro.

## 9.4. Safety

# 9.4.1. Hypoglycemia

Patients are encouraged to perform SMBG, whenever hypoglycemia may be suspected, either by symptoms experienced or perceived increased risk as related to dietary intake, physical activity, or inadvertent or atypical insulin dosing. All patients will be instructed to treat a BG  $\leq$ 70 mg/dL (3.9 mmol/L) as hypoglycemia.

Hypoglycemia events will be collected in eCOA (see Section 9.1.4.1). If a hypoglycemia event is suspected, the patient should record the BG value, any associated symptoms, and the treatment administered in eCOA. The patient should contact the site as necessary. Reports of hypoglycemia will be classified by the investigator as "severe" or "not severe" based upon data collected in eCOA and in consultation with the patient; see below and Section 9.2.1. All episodes of severe hypoglycemia must be reported as AEs via electronic data entry and as SAEs.

Hypoglycemia will be described using the following definitions:

#### Documented hypoglycemia:

- o **Documented symptomatic hypoglycemia:** an event during which typical symptoms of hypoglycemia are accompanied by BG ≤70 mg/dL (3.9 mmol/L).
- o **Documented asymptomatic hypoglycemia:** an event not accompanied by typical symptoms of hypoglycemia but with  $BG \le 70 \text{ mg/dL}$  (3.9 mmol/L).
- Documented unspecified hypoglycemia: an event during which BG ≤70 mg/dL (3.9 mmol/L) but no information relative to symptoms of hypoglycemia were recorded.
- **Probable symptomatic hypoglycemia:** an event during which symptoms are indicative of hypoglycemia and which was presumably caused by BG ≤70 mg/dL (3.9 mmol/L), although no BG measurement was reported.
- Severe hypoglycemia: an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. During these episodes, the patient has an altered mental status and cannot assist in his/her own care, may be semiconscious or unconscious, or experience coma with or without seizures, and may require parenteral therapy. BG measurements may not be available during such an event, but neurological recovery attributable to the restoration of BG concentration to normal is considered sufficient evidence that the event was induced by a low BG concentration (BG ≤70 mg/dL [3.9 mmol/L]).
- **Nocturnal hypoglycemia:** any hypoglycemic event (documented hypoglycemia or probable symptomatic hypoglycemia, including severe hypoglycemia) that occurs between bedtime and waking.
- **Relative hypoglycemia:** an event during which typical symptoms of hypoglycemia, that do not require the assistance of another person, are accompanied by BG >70 mg/dL (3.9 mmol/L), but these levels may be quickly approaching the 70 mg/dL (3.9 mmol/L) threshold.
- Overall hypoglycemia: This category combines all cases of hypoglycemia (documented hypoglycemia and probable symptomatic hypoglycemia, including

severe hypoglycemia) excluding the events of relative hypoglycemia. If an event of hypoglycemia falls into multiple subcategories, the event is only counted once in this category.

## 9.4.2. Severe Hypoglycemia

The determination of a hypoglycemic event as an episode of severe hypoglycemia as defined above, is made by the investigator based upon the medical need of the patient to have required assistance and is not predicated on the report of a patient simply having received assistance.

## 9.4.3. Electrocardiograms

For each patient, ECGs should be performed at Visit 1 according to the study-specific requirements described in the Schedule of Activities (Section 2).

ECGs will be interpreted by a qualified physician (the investigator or qualified designee) at the site as soon after the time of ECG collection as possible, and ideally while the patient is still present, to determine whether the patient meets entry criteria and for immediate patient management, should any clinically relevant findings be identified.

ECGs may be obtained at additional times, when deemed clinically necessary.

## 9.4.4. Vital Signs

For each patient, vital sign measurements should be conducted according to the Schedule of Activities (Section 2) including the study specific requirements.

# 9.4.5. Laboratory Tests

For each patient, laboratory tests detailed in Appendix 2 should be conducted according to the Schedule of Activities (Section 2 and Appendix 8).

Any clinically significant findings from laboratory tests that result in a diagnosis and that occur after the patient receives the first dose of IP should be reported to Lilly or its designee as an AE via electronic data entry.

# 9.4.6. Safety Monitoring

Lilly will periodically review evolving aggregate safety data within the study by appropriate methods.

If a study patient experiences elevated ALT  $\geq$ 3X ULN, ALP  $\geq$ 2X ULN, or elevated TBL  $\geq$ 2X ULN, clinical and laboratory monitoring should be initiated by the investigator. Details for hepatic monitoring depend upon the severity and persistence of observed laboratory test abnormalities. To ensure patient/patient safety and comply with regulatory guidance, the investigator is to consult with the Lilly CRP regarding collection of specific recommended clinical information and follow-up laboratory tests. See Appendix 4.

#### 9.5. Pharmacokinetics

Not applicable.

### 9.6. Pharmacodynamics

Not applicable.

## 9.7. Pharmacogenomics

# 9.7.1. Whole Blood Samples for Pharmacogenetic Research

A whole blood sample will be collected for pharmacogenetic analysis as specified in the Schedule of Activities (Section 2) where local regulations and ERBs allow.

Samples will not be used to conduct unspecified disease or population genetic research either now or in the future. Samples will be used to investigate variable response to LY900014 and to investigate genetic variants thought to play a role in T1D and related complications. Assessment of variable response may include evaluation of AEs or differences in efficacy.

All pharmacogenetic samples will be coded with the patient number. These samples and any data generated can be linked back to the patient only by the investigator site personnel. Samples will be destroyed according to a process consistent with local regulations.

Samples will be retained for a maximum of 15 years after the last patient visit for the study, or for a shorter period if local regulations and/or ERBs/institutional review boards impose shorter time limits, at a facility selected by Lilly or its designee. This retention period enables use of new technologies, response to regulatory questions, and investigation of variable response that may not be observed until later in the development of LY900014 or after LY900014 becomes commercially available.

Molecular technologies are expected to improve during the 15-year storage period and therefore cannot be specifically named. However, existing approaches include whole genome or exome sequencing, genome wide association studies, candidate gene studies, and epigenetic analyses. Regardless of technology utilized, genotyping data generated will be used only for the specific research scope described in this section.

# 9.8. Biomarkers and Predictive or Other Analyses

Serum and plasma samples for nonpharmacogenetic biomarker research will be collected at the times specified in the Schedule of Activities (Section 2) where local regulations allow.

Biomarker research is performed to address questions of relevance to drug disposition, target engagement, pharmacodynamics, mechanism of action, variability of patient response (including safety), and clinical outcome. Sample collection is incorporated into clinical studies to enable examination of these questions through measurement of biomolecules including DNA, RNA, proteins, lipids, and other cellular elements.

Samples will be used for research on the drug target, disease process, variable response to LY900014, pathways associated with T1D, mechanism of action of LY900014, and/or research method or in validating diagnostic tools or assay(s) related to T1D.

All samples will be coded with the patient number. These samples and any data generated can be linked back to the patient only by the investigator site personnel. Samples will be destroyed according to a process consistent with local regulations.

Samples will be retained for a maximum 15 years after the last patient visit for the study, or for a shorter period if local regulations and ERBs impose shorter time limits, at a facility selected by Lilly or its designee. This retention period enables use of new technologies, response to regulatory questions, and investigation of variable response that may not be observed until later in the development of LY900014 or after LY900014 become(s) commercially available.

## 9.8.1. Samples for Immunogenicity Testing

Blood samples for immunogenicity testing will be collected to determine antibody production against insulin lispro as specified in the Schedule of Activities (Section 2 and Appendix 8).

Immunogenicity will be assessed by a validated radio ligand-binding assay (RBA) to detect antiinsulin lispro antibodies in the presence of lispro. Instead of quantitating the level of anti-insulin lispro antibodies by titer, the RBA reports a semiquantitative percent-binding for each positive sample. Additionally, positive samples will be characterized for cross-reactive binding to native insulin.

Clinical and reliable on-market data indicate that the immunogenic potential of insulin lispro is comparable to other marketed insulins such as regular human insulin (Fineberg et al. 1996) and, when present, anti-insulin antibodies do not appear to be clinically consequential (Fineberg et al. 2003). Therefore, rather than relying on an in vitro neutralization assay, well established in vivo measures of insulin lispro efficacy (that is, insulin dose, HbA1c) will be utilized to directly monitor for any potential neutralizing effect of anti-lispro antibodies.

Patients who complete the 4-week safety follow-up visit and have treatment-emergent antiinsulin lispro antibodies that have not returned to prespecified baseline range (Visit 2) will be asked to participate in follow-up to monitor antibody levels. Instructions for this follow-up assessment are provided in Appendix 8.

Samples will be retained for a maximum of 15 years after the last patient visit for the study, or for a shorter period if regulations and ERBs impose shorter time limits, at a facility selected by Lilly or its designee. The duration allows the sponsor to respond to future regulatory requests related to LY900014.

#### 9.9. Health Economics

The self-reported questionnaires will be administered according to the Schedule of Activities (Section 2) in countries where the questionnaires have been translated into the native language of the region and linguistically validated.





## 9.9.2. Insulin Treatment Satisfaction Questionnaire

The Insulin Treatment Satisfaction Questionnaire (ITSQ) (Anderson et al. 2004) is a validated instrument containing 22 items that assesses treatment satisfaction for persons with diabetes on







### 10. Statistical Considerations

### 10.1. Sample Size Determination

Approximately 1199 patients will be randomized in order that 1020 patients complete the study through the primary endpoint at Week 26.

The primary objective of this study is to test the hypothesis that LY900014 is noninferior to insulin lispro on glycemic control as measured by change from baseline to Week 26 in HbA1c in patients with T1D when administered in a double-blind manner as prandial insulin (0-2 minutes before meals) in combination with basal insulin.

Patients will be randomized in a 4:4:3 ratio to double-blind LY900014 dosed 0 to 2 minutes before meals, double-blind insulin lispro dosed 0 to 2 minutes before meals, or open-label LY900014 dosed 20 minutes after the start of a meal (LY900014+20). Assuming a noninferiority margin (NIM) of 0.4%, no true difference between treatment arms, and an SD of 1.1%, approximately 371 completers in each double-blind treatment group will provide at least 99% power to show noninferiority between LY900014 and insulin lispro in change from baseline to 26 weeks in HbA1c using the upper limit of a 2-sided 95% confidence interval (CI) (LY900014 – insulin lispro). Assuming a 15% dropout rate for 26 weeks, approximately 1199 patients (436 in each double-blind treatment group and 327 in the open-label treatment group) will need to be randomized. This sample size also has 95% power to show noninferiority between LY900014 and insulin lispro using a 0.3% NIM at 26 weeks.

# 10.2. Populations for Analyses

For purposes of analysis, the following populations are defined:

| Population | Description |
|---|---|
| Entered | All patients who give informed consent. |
| Enrolled | All patients who receive at least 1 dose of open-label insulin lispro in the 8-week lead-in period. |
| Randomized | All patients who are randomly assigned to study treatment at Visit 8. Treatment group will be |
| | defined on the basis of the treatment the patients are assigned. |
| Safety | All randomized patients who receive at least 1 dose of the randomly assigned IP. |
| Completer | Patients included in the randomized population who have completed Week 26 of study treatment |
| | without permanent discontinuation of IP. |
| Per Protocol | Patients included in the randomized population who have completed Week 26 of study treatment |
| | without permanent discontinuation of IP and without significant protocol deviations through |
| | Week 26 that would significantly impact the primary objective. |
| | Treatment group will be defined on the basis of the treatment the patients actually receive. |

# 10.3. Statistical Analyses

#### 10.3.1. General Statistical Considerations

Statistical analysis of this study will be the responsibility of Lilly or its designee. Any change to the data analysis methods described in the protocol will require an amendment ONLY if it

changes a principal feature of the protocol. Any other change to the data analysis methods described in the protocol, and the justification for making the change, will be described in the statistical analysis plan (SAP) or the clinical study report (CSR). Additional exploratory analyses of data will be conducted, as deemed appropriate.

The primary analysis is for the treatment period through Week 26. The primary endpoint is the HbA1c measurement obtained at Week 26 (Visit 18). The measurement obtained at Week 52 (Visit 22) will be a secondary endpoint.

Efficacy analyses will be conducted on all randomized patients according to the treatment the patients are assigned. The analyses for the primary and multiplicity adjusted objectives will be performed for the efficacy estimand including data collected prior to permanent discontinuation of IP through Week 26 and for the ITT estimand (treatment regimen estimand) including all data collected through Week 26 regardless of IP use (Section 10.3.3.1). Unless otherwise specified, the efficacy analyses for other secondary objectives and exploratory objectives will be performed for the efficacy estimand. When change from baseline is included as a response variable of analysis models, the patient will be included in the analysis only if he/she has a baseline and a postbaseline measurement. Selected efficacy analyses will also be conducted using the Per-Protocol (PP) and Completer populations. Week 52 analyses will include the LY900014 and insulin lispro treatment and only be performed for the efficacy estimand.

Safety analyses will be conducted on the Safety population. Analyses of AEs will include 2 sets of analyses, unless otherwise specified. The first set of analyses will include data collected prior to permanent discontinuation of IP. The second set of analyses will include all data collected during the course of the entire study regardless of IP use. Analyses of hypoglycemia will be conducted on data collected prior to permanent discontinuation of IP, while analyses for post-treatment may be conducted as needed. Analyses of safety laboratory measurements will be performed on all data collected during the planned treatment period regardless of IP use. Week 26 analyses will include treatment comparisons among the three treatment groups. Week 52 analyses will also include data collected during the follow-up visit for LY900014 and insulin lispro. All data collected including the follow-up visit will be summarized for LY900014+20.

Unless otherwise noted, all tests of treatment effects will be conducted at a 2-sided alpha level of 0.05, and CIs will be calculated at 95%, 2-sided. All tests of interactions between treatment groups and other factors will be conducted at a 2-sided alpha level of 0.10. Countries in similar geographic regions with fewer than 10 patients, based on the all-randomized population, will be pooled to achieve a pooled country of at least 10 patients. All analyses using country in the model will use a pooled country, unless otherwise specified. The final pooling by country and geographic region will be finalized prior to data lock.

A graphical approach for multiple comparisons (Bretz et al. 2011) will be used to strongly control the overall Type I error (2-sided alpha level of 0.05) for testing the treatment effect for the primary and multiplicity adjusted objectives.

Baseline is defined as the last nonmissing measurement at or before the randomization visit, (Visit 8) unless otherwise specified.

A restricted maximum likelihood based, mixed-effect model repeated measure (MMRM) analysis will be used to analyze continuous longitudinal variables. All the longitudinal observations at each scheduled postbaseline visit will be included in the analysis. The model for the analysis of the primary efficacy endpoint of change from baseline in HbA1c will include the fixed class effects of treatment, strata (pooled country, type of basal insulin, and prandial insulin dosing plan), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariate of baseline value. For analyses of variables other than HbA1c, the HbA1c stratum (≤7.5%, >7.5%) will be included in the model. An unstructured covariance structure will be used to model the within-patient errors. Significance tests will be based on least squares (LS) means and Type III tests. SAS PROC MIXED will be used to perform the analysis. If this analysis fails to converge, the following covariance structures will be tested in order:

- Toeplitz with heterogeneity
- Autoregressive with heterogeneity
- Compound symmetry with heterogeneous variances
- Toeplitz
- Autoregressive
- Compound symmetry without heterogeneous variances.

The first covariance structure that converges will be used. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom.

Analysis of covariance (ANCOVA) will also be used to analyze continuous variables. The model for the change from baseline to the Week 26 HbA1c endpoint will include treatment and strata (pooled country, type of basal insulin, and prandial insulin dosing plan) as fixed effects and baseline as a covariate. Unless otherwise stated, missing endpoints will be imputed using the last-observation−carried-forward (LOCF) approach, using only postbaseline data. For analyses of variables other than HbA1c, the HbA1c stratum (≤7.5%, >7.5%) will be included in the model.

For continuous measures, summary statistics will include sample size, mean, SD, median, minimum, and maximum for both the actual and the change from baseline measurements. LS means and standard errors derived from the analysis models will also be displayed for the change from baseline measurements. Treatment comparisons will be displayed showing the treatment difference LS means and the 95% CIs for the treatment differences, along with the p-values for the treatment comparisons.

For categorical measures, summary statistics will include sample size, frequency, and percentages. Fisher's exact test or Pearson's chi-square test will be used for treatment comparisons.

### 10.3.2. Treatment Group Comparability

#### 10.3.2.1. Patient Disposition

A detailed description of patient disposition will be provided. Frequency counts and percentages of all patients entered, enrolled, randomized, completing, and/or discontinuing from the study will be presented for each treatment group. Reasons for discontinuation from study treatment and from the study during the treatment period will be summarized and compared between treatment groups using Fisher's exact tests. Reasons for discontinuation from the study during the lead-in and follow-up periods will be summarized.

#### 10.3.2.2. Patient Characteristics

Standard baseline characteristics of age, sex, ethnicity, race, height, weight, and BMI will be summarized for all randomized patients. Summary statistics will include sample size, mean, SD, median, minimum, and maximum for continuous measures and sample size, frequency, and percent for categorical measures. Comparisons between treatment groups will be performed using Fisher's exact test or Pearson's chi-square test for categorical data and an analysis of variance (ANOVA) with treatment in the model for continuous data. Baseline diabetes characteristics will be summarized in a similar manner.

Medical history and AEs at baseline will be summarized by preferred term (PT) within system organ class (SOC), and comparison between treatment groups will be performed using Fisher's exact test.

## 10.3.2.3. Concomitant Therapy

The type of insulin therapy at study entry and at baseline will be compared between treatment groups using Fisher's exact tests. The dose of basal and bolus insulin therapy during the lead-in period will be compared between treatment groups using an ANOVA with treatment in the model.

Concomitant medications used during the treatment period will be summarized and compared between treatment groups using Fisher's exact test.

## 10.3.2.4. Treatment Compliance

The proportions of patients compliant with timing of prandial insulin administration relative to meal time (premeal and postmeal) will be summarized.

# 10.3.3. Efficacy Analyses

## 10.3.3.1. Primary Analyses

The primary objective of this study is to test the hypothesis that LY900014 is noninferior to insulin lispro on glycemic control (NIM=0.4% for HbA1c) in patients with T1D, when administered as prandial insulin (0-2 minutes prior to the meal), in combination with basal insulin for 26 weeks. There will be 2 primary analysis methods, each tested at the full significance level of 0.05.

For the US FDA submission, the primary analysis method will use the copy reference approach to impute missing data based on multiple imputations with a pattern mixture model. This

analysis is for the ITT estimand that will include all data collected from randomization through Week 26, regardless of IP use. The reference will be all observed data from the randomized patients in the same treatment group who discontinue IP and complete the study without missing data. After imputation, the primary efficacy comparison will be based on the contrast between LY900014 and insulin lispro from the ANCOVA analysis of change from baseline to Week 26 in HbA1c using all randomized patients as described in Section 10.3.1.

If there are only a limited number of patients in the reference group as described above that leads to a failure in performing the proposed multiple imputation analysis, the reference will be changed to include all observed data from all randomized patients in the same treatment arm who complete the study without missing data.

For non-FDA submissions and publications, the primary efficacy comparison will be based on the contrast between LY900014 and insulin lispro at Week 26 (Visit 18) from the MMRM analysis of change from baseline in HbA1c including data collected from all randomized patients prior to permanent discontinuation of IP through Week 26 (efficacy estimand). The analysis model and selection of covariance structure are described in Section 10.3.1.

For both primary analysis approaches, LY900014 will be declared noninferior to insulin lispro if the upper limit of the 2-sided 95% CI for the LS mean difference in the change from baseline in HbA1c for LY900014 minus insulin lispro is below +0.4%. In addition, the 95% CI for the treatment difference will be compared to an alternative NIM of +0.3%. Both estimands will be tested at the full significance level of 0.05. The ANCOVA and MMRM analyses will include data from all 3 treatment groups; however, the contrasts between LY900014+20 and insulin lispro and between LY900014 and LY900014+20 are not part of the primary efficacy comparisons.

In addition to the primary objective, the superiority of LY900014 in controlling HbA1c compared to insulin lispro will also be assessed for each analysis approach described above. If the p-value is less than the alpha level from the graphical approach allocated to the superiority hypothesis, LY900014 will be declared superior to insulin lispro.

### 10.3.3.1.1. Sensitivity Analyses for Missing Data

A missing-not-at-random (MNAR)-based analysis will be performed for both the efficacy and ITT estimands to assess sensitivity to departures from the missing-at-random (MAR) assumption by repeatedly adjusting the imputations of missing data to provide a progressively more severe stress test (Ratitch et al. 2013). The basic idea is to impute the missing values and add a value (delta) to the imputed values of the experimental treatment group and perform an analysis for the primary endpoint on the delta-adjusted data set to see whether the conclusion of the primary analysis is overturned. If not, a larger delta is chosen and the process repeated until the primary result is overturned. If the delta required to overturn the primary result is not a plausible departure from MAR, then the primary result is robust to plausible departures from MAR. Imputation under the noninferiority null method (where delta equals the NIM) will be included as a special case of the progressive stress test.

For the ITT estimand, the reference group will be as described for the FDA primary analysis, and ANCOVA on the change from baseline to Week 26 in HbA1c will be used.

For the efficacy estimand, the reference group will be the insulin lispro treatment group. Imputation will be for all longitudinal visits

### 10.3.3.1.2. Additional Analyses for the Primary Endpoint

The primary MMRM analysis model will be repeated using the PP and Completer populations to check the sensitivity of the analysis. If the conclusion differs from that of all randomized patients, the data and analyses will be further investigated.

A secondary analysis model for the efficacy estimand will be an ANCOVA for HbA1c change from baseline to Week 26 (Visit 18), using the model described in Section 10.3.1. Missing endpoints will be imputed using the LOCF approach using postbaseline data only.

### 10.3.3.2. Secondary Analyses

A graphical approach for multiple comparisons will be used to strongly control the overall Type I error (2-sided alpha level of 0.05) for testing the treatment effect for the primary and the following multiplicity adjusted objectives: superiority of LY900014 compared with insulin lispro for 1-hour PPG excursion at Week 26, 2-hour PPG excursion at Week 26, and change from baseline to Week 26 in HbA1c; and noninferiority of LY900014+20 to insulin lispro in change from baseline to Week 26 in HbA1c. Analyses will be performed for both the efficacy estimand and ITT estimand as described in Section 10.3.3.1 using the same graphical testing scheme.

The graphical testing scheme will be described in the SAP. The study total alpha level (or study-wise type I error) is preset to be 5% for each estimand. The study total alpha level will be used for the primary objective in the initial step. The alpha level will be allocated to other key endpoints based on the weights in testing paths once the primary endpoint is successfully demonstrated. If 1 of the remaining hypotheses is successfully demonstrated with the preserved alpha level, its preserved alpha will be allocated to the remainder of the hypotheses by the weights in the paths. The iterative test procedure continues until none of the remaining hypotheses can be demonstrated with their preserved alphas or all hypotheses are demonstrated successful.

An ANCOVA model with strata (pooled country, type of basal insulin, prandial insulin dosing plan, and baseline HbA1c strata [(≤7.5%, >7.5%]) and treatment as fixed effects and baseline as a covariate will be used to analyze the 1-hour and 2-hour PPG excursions. However, if the percentage of the patients with missing MMTT data at baseline is higher than 15%, a constrained longitudinal data analysis model (Liu et al. 2009; Lu 2010) will be used instead. Analyses details will be documented in the SAP.

Superiority in change from baseline in HbA1c for LY900014 compared with insulin lispro and noninferiority in change from baseline in HbA1c for LY900014+20 to insulin lispro will be determined from the analysis approaches outlined in Section 10.3.3.1

HbA1c and change from baseline in HbA1c at all time points will be analyzed by the same MMRM model used for the primary analysis for the efficacy estimand.

Additional continuous secondary efficacy variables, as well as the change from baseline for these variables, will be analyzed either by the MMRM or ANCOVA models described in Section 10.3.1 for the efficacy estimand.

Treatment comparisons for the proportion of patients with HbA1c <7.0% and  $\leq$ 6.5% will be analyzed using a longitudinal logistic regression with repeated measurements conducted by a generalized linear mixed model including independent variables of treatment, baseline HbA1c value, visit, baseline HbA1c by visit interaction, and treatment by visit interaction. An unstructured covariance structure will be used. As a sensitivity analysis, the proportion of patients with HbA1c <7.0% and  $\leq$ 6.5% at Week 26 (Visit 18), imputed using LOCF, will be compared using a logistic regression model including treatment and baseline HbA1c value in the model.

Actual and change from baseline in basal, prandial, and total dose, as well as the prandial/total insulin dose ratio, will be analyzed by the MMRM models described in Section 10.3.1.

Analyses of efficacy data collected from randomization through Week 52 for comparisons of the LY900014 and insulin lispro treatment groups will be similar to those described above for the efficacy estimand.

### 10.3.3.3. Tertiary/Exploratory Analyses

Continuous variables and the change from baseline for these variables will be analyzed either by the MMRM or ANCOVA models described in Section 10.3.1. Categorical variables will be analyzed either by model (for example, logistic regression) or by Fisher's exact test or Pearson's chi-square test. Analysis details for the tertiary endpoints will be described in the SAP.

# 10.3.4. Safety Analyses

Safety measures will include AEs, hypoglycemia, vital signs and weight, treatment exposure, laboratory measures, and antibodies to insulin lispro. Analyses will be performed on data collected from randomization through Week 26 for all 3 treatment groups and for data collected from randomization through Week 52 for the LY900014 and insulin lispro treatment groups.

Events that are newly reported after the first dose of IP or reported to worsen in severity from baseline will be considered treatment-emergent AEs (TEAEs). The Medical Dictionary for Regulatory Activities (MedDRA) lowest level term (LLT) will be used in the treatment-emergent assessment. The maximum severity for each LLT during the baseline period will be used as baseline severity.

SAEs, AEs reported as reason for discontinuation from the IP or study, and TEAEs will be summarized in tables using the MedDRA PT, sorted by decreasing frequency within the LY900014 treatment group. TEAEs will also be summarized by PT sorted by decreasing frequency within SOC for all TEAEs and by maximum severity. For events that are specific to only one sex, the denominator and computation of the percentage will include only patients from

the given sex. The number and proportion of patients with at least 1 event for each type of event will be summarized and compared between treatment groups using Fisher's exact test. SAEs, AEs reported as reason for discontinuation from the study, and TEAEs will also be summarized for open-label insulin lispro during the lead-in period.

Hypoglycemia rates will be summarized for periods of 30 days, 1 year, and 100 years (severe hypoglycemia only). The rate of severe hypoglycemia per 100 years will be compared between treatment groups using the empirical method (details will be described in SAP). For each of the other categories of hypoglycemia, the number of hypoglycemia events during a specific period (rate) after randomization (for example, Weeks 0-12 of treatment period) will be analyzed by using a negative binomial regression model. The model will include treatment and the baseline hypoglycemia rate (measured during lead-in) as a covariate. An offset defined as the log transformation of treatment exposure in the specific period (days)/365.25 days (or 30 days) will be included in the model to estimate the rate of hypoglycemia per year (or per 30 days). The proportion of patients with at least 1 hypoglycemic event in each category (incidence) during a specific period after randomization will be analyzed using a logistic regression model including treatment and baseline hypoglycemia rate value in the model.

Continuous safety variables, as well as the change from baseline for these variables, will be analyzed by MMRM or ANCOVA models. For categorical variables, Fisher's exact test or Pearson's chi-square test will be used to compare treatment groups unless otherwise specified.

The analyses for assessing immunogenicity data will be described in the SAP after being agreed with the FDA on the threshold for determining treatment-emergent antibodies to insulin lispro.

# 10.3.5. Other Analyses



For the ITSQ, the change from baseline to LOCF endpoint while on treatment in each domain transformed score (inconvenience, lifestyle, hypoglycemic control, glycemic control, delivery system) and overall transformed score will be analyzed using the ANCOVA model described in Section 10.3.1.



Analyses of health economics data collected from randomization through Week 52 for comparisons of the LY900014 and insulin lispro treatment groups will be similar to those described above.

### 10.3.5.2. Subgroup Analyses

The following subgroups will be analyzed using the efficacy estimand to evaluate consistency of treatment effects on the primary efficacy measure if there are sufficient numbers of patients in each treatment by subgroup (for example, 10%):

- Age (<40 years,  $\ge40$  years)
- HbA1c stratum ( $\leq 7.5\%$ , > 7.5%)
- Type of basal insulin during the lead-in period (glargine U-100, degludec U-100)
- Prandial insulin dosing plan (carbohydrate counting, pattern adjustment)
- Patient's personal CGM/FGM use during the study (Yes, No)
- Sex (male or female)
- BMI (<25,  $\ge 25$  kg/m<sup>2</sup> and <30,  $\ge 30$  kg/m<sup>2</sup>)
- Duration of diabetes (using the median as the cut-off)
- Race
- Ethnicity
- Country
- Region
- Baseline 1-hour PPG excursion
- Baseline 1-hour PPG (PPG  $\leq$ 180 mg/dL,  $\geq$ 180 mg/dL)
- Baseline 2-hour PPG excursion
- Baseline 2-hour PPG (PPG ≤180 mg/dL, >180 mg/dL)

Analyses for HbA1c and change from baseline in HbA1c will be performed using an MMRM model that includes the same fixed effects given for the primary analysis model plus factors of subgroup, 2-way interaction of subgroup and treatment, 2-way interaction of subgroup and visit, and 3-way interaction of treatment, visit and subgroup. The interaction of subgroup and treatment at the primary endpoint (Week 26) will be evaluated to assess the treatment by subgroup interaction. When analyzing HbA1c stratum (≤7.5%, >7.5%) as a subgroup, the baseline HbA1c will be not be included as a covariate to avoid confounding.

Additional subgroup analyses may also be performed.

# 10.3.6. Interim Analyses

No interim analyses are planned for this study. If an unplanned interim analysis is deemed necessary, the appropriate Lilly medical director, or designee, will be consulted to determine whether it is necessary to amend the protocol.

The primary database lock will occur after all patients in the double-blind arms have either completed the Week 26 visit or discontinued from the study prior to Week 26, and after all patients in the open-label treatment group have completed Visit 801. Investigators and patients will remain blinded to treatment assignments until the final database lock after all patients

complete the study as described in Section 7.3. Unblinding details are specified in the unblinding plan section of the SAP or a separate unblinding plan document.

### 11. References

- Alberti KG, Zimmet PZ. Definition, diagnosis and classification of diabetes mellitus and its complications. Part 1: diagnosis and classification of diabetes mellitus provisional report of a WHO consultation. *Diabet Med.* 1998;15(7):539-553.
- Anderson RT, Skovlund SE, Marrero D, Levine DW, Meadows K, Brod M, Balkrishnan R. Development and validation of the insulin treatment satisfaction questionnaire. *Clin Ther*. 2004;26(4):565-578.
- Bailey TS, Grunberger G, Bode BW, Handelsman Y, Hirsch IB, Jovanovič L, Roberts VL, Rodbard D, Tamborlane WV, Walsh J; American Association of Clinical Endocrinologists (AACE); American College of Endocrinology (ACE). American Association of Clinical Endocrinologists and American College of Endocrinology 2016 outpatient glucose monitoring consensus statement. *Endocr Pract*. 2016;22(2):231-261.
- Barrett KE, Barman SM, Boitano S, Brooks HL. Ganong's review of medical physiology. 25th ed. New York: McGraw-Hill Education; 2016. Chapter 24.
- Bartley PC, Bogoev M, Larsen J, Philotheou A. Long-term efficacy and safety of insulin detemir compared to Neutral Protamine Hagedorn insulin in patients with Type 1 diabetes using a treat-to-target basal-bolus regimen with insulin aspart at meals: a 2-year, randomized, controlled trial. *Diabet Med.* 2008;25(4):442-449.
- Bennett P. Classification and diagnosis of diabetes mellitus and impaired glucose tolerance. In: Pickup JC, William G, editors. Textbook of diabetes. Vol. 1. 1st ed. Oxford: Blackwell Scientific Publications; 1991:p 37-44.
- Bergenstal RM, Johnson M, Powers MA, Wynne A, Vlajnic A, Hollander P, Rendell M. Adjust to target in type 2 diabetes: comparison of a simple algorithm with carbohydrate counting for adjustment of mealtime insulin glulisine. *Diabetes Care*. 2008;31(7):1305-1310.
- Bolli GB, Kerr D, Thomas R, Torlone E, Sola-Gazagnes S, Vitacolonna E, Selam JL, Home PD. Comparison of a multiple daily insulin injection regime (basal once-daily glargine plus mealtime lispro) and continuous subcutaneous insulin infusion (lispro) in type 1 diabetes: a randomized open parallel multicenter study. *Diabetes Care*. 2009;32(7):1170-1176. Erratum in: *Diabetes Care*. 2009;32(10):1944.
- Bretz F, Posch M, Glimm E, Klinglmueller F, Maurer W, Rohmeyer K. Graphical approaches for multiple comparison procedures using weighted Bonferroni, Simes, or parametric tests. *Biom J.* 2011;53(6):894-913.
- Fineberg NS, Fineberg SE, Anderson JH, Birkett MA, Gibson RG, Hufferd S. Immunologic effects of insulin lispro [Lys (B28), Pro (B29) human insulin] in IDDM and NIDDM patients previously treated with insulin. *Diabetes*. 1996;45(12):1750-1754.
- Fineberg SE, Huang J, Brunelle R, Gulliya KS, Anderson JH Jr. Effect of long-term exposure to insulin lispro on the induction of antibody response in patients with type 1 or type 2 diabetes. *Diabetes Care*. 2003;26(1):89-96.
- Gan MJ, Albanese-O'Neill A, Haller MJ. Type 1 diabetes: current concepts in epidemiology, pathophysiology, clinical care, and research. *Curr Probl Pediatr Adolesc Health Care*. 2012:42(10):269-291.
- Humalog [package insert]. Indianapolis, IN: Eli Lilly and Company; 2015.
- Humalog [summary of product characteristics]. The Netherlands. Eli Lilly Nederland B.V; 2016.
- Liu GF, Lu K, Mogg R, Mallick M, Mehrotra DV. Should baseline be a covariate or dependent variable in analyses of change from baseline in clinical trials? *Stat Med*. 2009;28(20):2509-2530.
- Lu K. On efficiency of constrained longitudinal data analysis versus longitudinal analysis of covariance. *Biometrics*. 2010;66(3):891-896.
- Monnier L, Lapinski H, Colette C. Contributions of fasting and postprandial plasma glucose increments to the overall diurnal hyperglycemia of type 2 diabetic patients: variations with increasing levels of HbA(1c). *Diabetes Care*. 2003;26(3):881-885.
- [PMR] Pharmaceutical and healthcare market in CEE and CIS. Remodulin approved in 22 European countries, also Poland. PMR web site. Available at http://www.ceepharma.com/news/25318/remodulin-approved-in-22-european-countries-also-poland. Published September 1, 2005. Accessed September 16, 2016.
- Ratitch B, O'Kelly M, Tosiello R. Missing data in clinical trials: from clinical assumptions to statistical analysis using pattern mixture models. *Pharm Stat.* 2013;12(6):337-347.
- Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. *Pharmacoeconomics*. 1993;4(5):353-365.
- Remodulin [package insert]. Research Triangle Park, NC: United Therapeutics Corp; 2014.
- Scheiner G. Insulin-to-carb ratios made easy. Available at: http://integrateddiabetes.com/Articles/insu/carb%20ratio%20article%20for%20mendosa.pdf. Published November 2007. Accessed September 23, 2016.
- Stark Casagrande S, Fradkin JE, Saydah SH, Rust KF, Cowie CC. The prevalence of meeting A1C, blood pressure, and LDL goals among people with diabetes, 1988-2010. *Diabetes Care*. 2013;36(8):2271-2279.
- van Reenen M, Janssen B for the EuroQol Research Foundation. EQ-5D-5L User Guide: Basic information on how to use the EQ-5D-5L instrument. Available at: http://www.euroqol.org/fileadmin/user\_upload/Documenten/PDF/Folders\_Flyers/EQ-5D-5L\_UserGuide\_2015.pdf. Accessed December 12, 2016

# 12. Appendices

# Appendix 1. Abbreviations and Definitions

| Term | Definition |
|---|---|
| 1,5-AG | 1,5-Anhydroglucitol |
| AE | adverse event: Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| ANOVA | analysis of variance |
| AST | aspartate aminotransferase |
| BG | blood glucose |
| blinding/masking | A single-blind study is one in which the investigator and/or his staff are aware of the treatment but the patient is not, or vice versa, or when the sponsor is aware of the treatment but the investigator and/his staff and the patient are not. |
| | A double-blind study is one in which neither the patient nor any of the investigator or sponsor staff who are involved in the treatment or clinical evaluation of the patients are aware of the treatment received. |
| ВМІ | body mass index |
| CF | correction factor |
| CGM | continuous glucose monitoring |
| CI | confidence interval |
| Product complaint | Product complaints are a customer's written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness, or performance of a Lilly product after it is released for distribution. |
| CRP/CRS | clinical research physician: Individual responsible for the medical conduct of the study. Responsibilities of the CRP may be performed by a physician, clinical research scientist, global safety physician, or other medical officer. |
| CSII | continuous subcutaneous insulin infusion |
| CSR | clinical study report |

ECG electrocardiogram

eCOA electronic clinical outcomes assessment

eCRF electronic case report form

enroll The act of assigning a patient to a treatment. Patients who are enrolled in the trial are those

who have been assigned to a treatment.

enter Patients entered into a trial are those who sign the informed consent form directly or through

their legally acceptable representatives.

# CCI

ERB ethical review board

FBG fasting blood glucose

FDA Food and Drug Administration

FGM flash glucose monitoring

GCP good clinical practice

GD glucodynamic(s)

GRAS Generally Recognized As Safe

HbA1c hemoglobin A1c

IB Investigator's Brochure

ICF informed consent form

ICH International Conference on Harmonisation

ICR insulin to carbohydrate ratio

IP investigational product: A pharmaceutical form of an active ingredient or placebo being

tested or used as a reference in a clinical trial, including products already on the market when used or assembled (formulated or packaged) in a way different from the authorized form, or marketed products used for an unauthorized indication, or marketed products used to gain

further information about the authorized form.

ITSQ Insulin Treatment Satisfaction Questionnaire

ITT intention to treat: The principle that asserts that the effect of a treatment policy can be best

assessed by evaluating on the basis of the intention to treat a patient (that is, the planned treatment regimen) rather than the actual treatment given. It has the consequence that patients allocated to a treatment group should be followed up, assessed, and analyzed as members of

that group irrespective of their compliance to the planned course of treatment.

IV intravenous

**IWRS** interactive web-response system

**LLT** lowest level term

**LOCF** last observation carried forward

**LS** least squares

MAR missing at random

MDI multiple daily injections

Medical Dictionary for Regulatory Activities

MMRM mixed-effect model repeated measure

MMTT mixed-meal tolerance test

**NIM** noninferiority margin

**NPH** neutral protamine Hagedorn

**PK** pharmacokinetic(s)

**PP** per protocol

**PPG** postprandial glucose

**PT** preferred term

**RBA** radio ligand-binding assay

**SAE** serious adverse event

**SAP** statistical analysis plan

SC Subcutaneous

**Screen** The act of determining if an individual meets minimum requirements to become part of a pool

of potential candidates for participation in a clinical study.

**SD** standard deviation

**SMBG** self-monitored blood glucose

**SOC** system organ class

**SUSARs** suspected unexpected serious adverse reactions

**T1D** type 1 diabetes

T2D type 2 diabetes

TBL total bilirubin level

TEADA treatment-emergent anti-insulin lispro antibody

TEAE treatment-emergent adverse event: An untoward medical occurrence that emerges during a

defined treatment period, having been absent pretreatment, or worsens relative to the

pretreatment state, which and does not necessarily have to have a causal relationship with this

treatment.

ULN upper limit of normal

URI ultra-rapid insulin

VAS visual analog scale



#### **Clinical Laboratory Tests** Appendix 2.

#### Clinical Laboratory Testsa

**Clinical Chemistry(Serum Concentrations of):** Hematology

Hemoglobin Sodium Hematocrit Potassium Erythrocyte count (RBC) Total bilirubin Mean cell volume Direct bilirubin Mean cell hemoglobin concentration Alkaline phosphatase

Leukocytes (WBC) Alanine aminotransferase (ALT) Neutrophils, segmented Aspartate aminotransferase (AST)

Lymphocytes Blood urea nitrogen (BUN)

Monocytes Creatinine Uric acid Eosinophils **Basophils** Calcium **Platelets** Chloride Magnesium

Urinalysis Total protein Specific gravity Glucose рН Albumin

Protein Creatine kinase (CK)

Glucose

Serum glucose, fasting Ketones Blood 1,5 Anhydroglucitol

Urine leukocyte esterase HbA1c

Bilirubin

Nitrite **Lipid Panel** LDLd

HDL

Serology Anti-insulin lispro antibodies Total cholesterol

**Triglycerides** 

Pregnancy Test (females only)b

Follicle-stimulating hormonec **Stored Samples** 

Pharmacogenetic samples

Nonpharmacogenetic biomarker samples

Abbreviations: HDL = high-density lipoproteins; IP = investigational product; LDL = low-density lipoproteins; RBC = red blood cells; WBC = white blood cells.

a All laboratory tests will be assayed by a Lilly-designated central laboratory, unless otherwise noted.

- b Serum pregnancy test must be performed in women of childbearing potential at Visit 1 followed by a urine pregnancy test within 24 hours prior to IP exposure at randomization and at other times at the investigator's discretion. When required per local regulations and/or institutional guidelines, local pregnancy testing will occur at mandatory times during the study treatment period.
- c Follicle-stimulating hormone test must be performed at Visit 1 for a postmenopausal woman who is between 50 and 54 years of age (inclusive) with an intact uterus, not on hormone therapy, and who has had at least 6 months of spontaneous amenorrhea.
- d This value will be calculated. If triglycerides >400 mg/dL, then direct LDL will be assayed.

# Appendix 3. Study Governance Considerations

# Appendix 3.1. Regulatory and Ethical Considerations, Including the Informed Consent Process

# Appendix 3.1.1. Informed Consent

The investigator is responsible for ensuring:

- that the patient understands the potential risks and benefits of participating in the study
- that informed consent is given by each patient or legal representative. This includes obtaining the appropriate signatures and dates on the ICF prior to the performance of any protocol procedures and prior to the administration of IP.
- answering any questions the patient may have throughout the study and sharing in a timely manner any new information that may be relevant to the patient's willingness to continue his or her participation in the trial.

# Appendix 3.1.2. Ethical Review

The investigator or an appropriate local representative must give assurance that the ERB was properly constituted and convened as required by International Conference on Harmonisation (ICH) guidelines and other applicable laws and regulations.

Documentation of ERB approval of the protocol and the ICF must be provided to Lilly before the study may begin at the investigative site(s). Lilly or its representatives must approve the ICF, including any changes made by the ERBs, before it is used at the investigative site(s). All ICFs must be compliant with the ICH guideline on GCP.

The study site's ERB(s) should be provided with the following:

- the current IB and updates during the course of the study
- ICF
- relevant curricula vitae

# Appendix 3.1.3. Regulatory Considerations

This study will be conducted in accordance with:

- consensus ethics principles derived from international ethics guidelines, including the Declaration of Helsinki and Council for International Organizations of Medical Sciences (CIOMS) International Ethical Guidelines
- applicable ICH GCP Guidelines
- applicable laws and regulations

Some of the obligations of the sponsor will be assigned to a third-party.

## Appendix 3.1.4. Investigator Information

Physicians with a specialty in endocrinology or primary care physicians specializing in endocrinology or internal medicine will participate as investigators in this clinical trial.

# Appendix 3.1.5. Protocol Signatures

The sponsor's responsible medical officer will approve the protocol, confirming that, to the best of his or her knowledge, the protocol accurately describes the planned design and conduct of the study.

After reading the protocol, each principal investigator will sign the protocol signature page and send a copy of the signed page to a Lilly representative.

## Appendix 3.1.6. Final Report Signature

The CSR coordinating investigator will sign the final CSR for this study, indicating agreement that, to the best of his or her knowledge, the report accurately describes the conduct and results of the study.

An investigator will be selected by the Lilly study team to serve as the CSR coordinating investigator. The sponsor's responsible medical officer and statistician will approve the final CSR for this study, confirming that, to the best of his or her knowledge, the report accurately describes the conduct and results of the study.

# Appendix 3.2. Data Quality Assurance

To ensure accurate, complete, and reliable data, Lilly or its representatives will do the following:

- provide instructional material to the study sites, as appropriate
- sponsor start-up training to instruct the investigators and study coordinators. This training will give instruction on the protocol, the completion of the case report forms (CRFs), and study procedures.
- make periodic visits to the study site
- be available for consultation and stay in contact with the study site personnel by mail, telephone, and/or fax
- review and evaluate CRF data and use standard computer edits to detect errors in data collection
- conduct a quality review of the database.

In addition, Lilly or its representatives will periodically check a sample of the patient data recorded against source documents at the study site. The study may be audited by Lilly or its representatives, and/or regulatory agencies at any time. Investigators will be given notice before an audit occurs.

The investigator will keep records of all original source data. This might include laboratory tests, medical records, and clinical notes. If requested, the investigator will provide the sponsor,

applicable regulatory agencies, and applicable ERBs with direct access to original source documents.

# Appendix 3.2.1. Data Capture System

An electronic data capture system will be used in this study. The site maintains a separate source for the data entered by the site into the sponsor-provided electronic data capture system.

Electronic clinical outcomes assessment (eCOA) measures (for example, a rating scale) or other data reported directly by the patient (for example, daily dosing schedule, event diary) are entered into an eCOA instrument (for example, personal digital assistant) at the time that the information is obtained. In these instances where there is no prior written or electronic source data at the site, the eCOA instrument record will serve as the source.

If eCOA records are stored at a third party site, investigator sites will have continuous access to the source documents during the study and will receive an archival copy at the end of the study for retention.

Any data for which the eCOA instrument record will serve to collect source data will be identified and documented by each site in that site's study file.

CRF data will be encoded and stored in a clinical trial database. Data managed by a central vendor, such as laboratory test data, will be stored electronically in the central vendor's database system. Data will subsequently be transferred from the central vendor to the Lilly data warehouse.

Data from complaint forms submitted to Lilly will be encoded and stored in the global product complaint management system.

# Appendix 3.3. Study and Site Closure

# Appendix 3.3.1. Discontinuation of Study Sites

Study site participation may be discontinued if Lilly, the investigator, or the ERB of the study site judges it necessary for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and GCP.

# Appendix 3.3.2. Discontinuation of the Study

The study will be discontinued if Lilly judges it necessary for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and GCP.

# Appendix 4. Hepatic Monitoring Tests for Treatment-Emergent Abnormality

Selected tests may be obtained in the event of a treatment-emergent hepatic abnormality and may be required in follow-up with patients in consultation with the Lilly, or its designee, clinical research physician.

| Hepatic | Mo | nitorir | ng Tests |
|---------|----|---------|----------|
|---------|----|---------|----------|

| Hepatic Hematologya | Haptoglobin <sup>a</sup> |
|---|---|
| Hemoglobin | |
| Hematocrit | Hepatic Coagulationa |
| RBC | Prothrombin time |
| WBC | Prothrombin time, INR |
| Neutrophils, segmented | |
| Lymphocytes | Hepatic Serologies <sup>a,b</sup> |
| Monocytes | Hepatitis A antibody, total |
| Eosinophils | Hepatitis A antibody, IgM |
| Basophils | Hepatitis B surface antigen |
| Platelets | Hepatitis B surface antibody |
| | Hepatitis B core antibody |
| Hepatic Chemistry <sup>a</sup> | Hepatitis C antibody |
| Total bilirubin | Hepatitis E antibody, IgG |
| Direct bilirubin | Hepatitis E antibody, IgM |
| Alkaline phosphatase | |
| ALT | Anti-nuclear antibodya |
| AST | |
| GGT | Alkaline phosphatase isoenzymesa |
| CPK | • |
| | Anti-smooth muscle antibody (or anti-actin antibody)a |

Abbreviations: ALT = alanine aminotransferase; AST = aspirate aminotransferase; CPK = creatinine phosphokinase; GGT = gamma-glutamyl transferase; Ig = immunoglobulin; INR = international normalized ratio; RBC = red blood cells; WBC = white blood cells.

- a Assayed by Lilly-designated or local laboratory (if test results are required urgently to manage patient care).
- b Reflex/confirmation dependent on regulatory requirements and/or testing availability.



# Appendix 6. New York Heart Association Cardiac Disease Classification

# **Functional Capacity**

#### Class I

Patients with cardiac disease but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain.

#### **Class II**

Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.

#### **Class III**

Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain.

#### Class IV

Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort increases.

1994 Revisions to Classification of Functional Capacity and Objective Assessment of Patients with Diseases of the Heart

www.americanheart.org. ©2011, American Heart Association, Inc.

# Appendix 7. Classification of Contraceptive Methods

Women of childbearing potential must use either 1 highly effective method of contraception or a combination of 2 effective methods of contraception. The patient may choose to use a double-barrier method of contraception (see chart below).

Barrier protection methods without concomitant use of a spermicide are not an effective
or acceptable method of contraception. Thus, each barrier method must include use of a
spermicide (that is, condom with spermicide, diaphragm with spermicide, female condom
with spermicide). It should be noted, however, that the use of male and female condoms
as a double-barrier method is not considered acceptable due to the high failure rate when
these barrier methods are combined.

## **Methods of Contraception**

| Highly Effective Methods of Contraception | Effective Methods of Contraception (must use combination of 2 methods) |
|---|---|
| Combined oral contraceptive pill and mini-pill | Male condom with spermicide |
| NuvaRing® | Female condom with spermicide |
| Implantable contraceptives | Diaphragm with spermicide |
| • Injectable contraceptives (such as Depo-Provera®) | Cervical sponge |
| • Intrauterine device (such as Mirena® and ParaGard®) | <ul> <li>Cervical cap with spermicide</li> </ul> |
| • Contraceptive patch – ONLY women <198 lb or 90 kg | |
| Total abstinence | |
| Vasectomy | |

# Appendix 8. Insulin Lispro Antibody Follow-Up Assessment

#### Rationale for Insulin Lispro Antibody Follow Up Assessment

As requested by the US FDA, any patient who develops a treatment-emergent anti-insulin lispro antibody (TEADA) response at any time during the study that has not returned to baseline by the completion of Visit 801 should undergo follow-up for antibodies to insulin lispro. Specific thresholds for determining treatment-emergent and return-to-baseline will be specified and documented in the SAP after being agreed with the FDA. Data collected during the insulin lispro antibody follow-up period is intended to evaluate whether antibodies to insulin lispro return to the prespecified baseline range and, in cases where antibodies remain elevated, to assess the possibility of loss of efficacy that may result from insulin neutralizing antibodies.

### Eligibility for Insulin Lispro Antibody Follow-Up Assessment

Any patient who develops a TEADA response that has not returned to the prespecified baseline range (based on Visit 2 sample) by the 4-week safety follow-up visit (based on Visit 801 sample) will undergo additional insulin lispro antibody monitoring. Study visits will continue at approximately 3-month intervals for a maximum of 6 months (approximately 26 weeks) after Visit 801 or until insulin lispro antibodies return to baseline range, whichever occurs sooner.

This follow-up assessment also includes any randomized patient who discontinues study insulin treatment prior to the end of the planned treatment period and has a TEADA response that has not returned to baseline range by Visit 801.

At Visit 801, it is recommended that the first insulin lispro antibody follow-up visit (Visit 802) be scheduled for <u>all</u> study patients, regardless of TEADA status. Visit 802 should occur approximately 13 weeks after Visit 801. Insulin lispro antibody percent binding results will not be provided to sites. When insulin antibody results are available, to determine whether the patient's insulin antibody levels have returned to baseline range, investigators will be notified and Visit 802 can be confirmed or cancelled as appropriate.

During the insulin lispro antibody follow-up period, investigators will be notified if insulin lispro antibodies for a given patient have returned to baseline range, at which time the patient's participation in the follow-up period should be stopped. In the exceptional circumstance that insulin antibody results are not available prior to the next scheduled follow-up visit, patients should be instructed to complete the visit as scheduled; however, the blood sample collected as part of the visit will only be analyzed if the insulin antibody results from the previous visit are still above baseline.

In any case, even where insulin antibodies persist, the insulin lispro antibody follow-up assessment is expected to last no longer than 30 weeks from the protocol-scheduled last treatment visit.

Patients should not participate in other clinical trials during the follow-up period. Patients entering the protocol as part of a maximized extended enrollment addendum (I8B-MC-ITRM[2]) will not be included in the insulin lispro antibody follow-up assessment.

#### Procedures for Insulin Lispro Antibody Follow-Up Assessment

In order to reduce potential interference with antibody monitoring during this follow-up period, introduction of new insulin formulations should be avoided. Guidance for diabetes therapy during the insulin antibody follow-up period is provided in Section 7.8.2.

Blood samples for insulin lispro antibody and HbA1c measurements should be collected at approximately 3-month intervals for up to 26 weeks after Visit 801. All SAEs (including severe hypoglycemia) and all nonserious AEs should be reported. Vital signs, body weight, total daily prandial insulin dose, total daily basal insulin dose, and information on concomitant medications will be collected at each insulin antibody follow-up visit as described in the Insulin Lispro Antibody Follow- Up Assessment Schedule of Activities (see chart below).

# Schedule of Activities during Insulin Lispro Antibody Follow-Up Assessment

| Study Period | Insulin Lispi<br>Follow-U | ED-IA<br>Follow-<br>Up | |
|---|---|---|---|
| eCRF Visit Number | 802 | 803 | |
| Visit Window (days) | ±14 | ±14 | |
| Time on Study Relative to Last Treatment Dose Visit (weeks) | 17 | 30 | |
| Time on Study Relative to First Treatment Dose Visit (weeks) | Open Label, 43 Double Blind, 69 | 56<br>82 | |
| IWRS | X | X | X |
| Dispense glucose monitoring and ancillary supplies | X | | |
| Telephone call for visit reminder or informing patient of completion in the study | X | X | |
| Return of unused diabetes medications and study supplies if required by local regulations | X | X | X |
| Concomitant medication | X | X | X |
| Total daily prandial insulin dose | X | X | X |
| Total daily basal insulin dose | X | X | X |
| Vital signs | X | X | X |
| Body weight | X | X | X |
| Adverse events and product complaints | X | X | X |
| Anti-insulin lispro antibodies | X | X | Xa |

Abbreviations: eCRF = electronic case report form; ED-IA = early discontinuation-insulin antibody; HbA1c = hemoglobin A1c; IWRS = interactive web response system.

X

HbA1c

<sup>&</sup>lt;sup>a</sup> Insulin lispro antibody samples collected as part of the ED-IA follow-up visit will be analyzed only if the results from the previous visit are still above baseline.

Appendix 9. Clinical Protocol Amendment I8B-MC-ITRM(a) Summary A Prospective, Randomized, Double-Blind Comparison of LY900014 to Insulin Lispro with an Open-Label Postprandial LY900014 Treatment Group, in Combination with Insulin Glargine or Insulin Degludec, in Adults with Type 1 Diabetes PRONTO-T1D

# **Overview**

Protocol I8B-MC-ITRM A Prospective, Randomized, Double-Blind Comparison of LY900014 to Insulin Lispro with an Open-Label Postprandial LY900014 Treatment Group, in Combination with Insulin Glargine or Insulin Degludec, in Adults with Type 1 Diabetes PRONTO-T1D has been amended. The new protocol is indicated by amendment (a) and will be used to conduct the study in place of any preceding version of the protocol.

The overall changes and rationale for the changes made to this protocol are described in the following table:

# Amendment Summary for Protocol I8B-MC-ITRM Amendment (a)

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Several Sections | Removed 'immediately following the meal, or whichevercomes first' LY900014 +20 arm will be 20 minutes after the start of the meal | In response to feedback from the FDA, the timing of postprandial administration of LY900014 was specified as 20 minutes after the start of the meal in order to ensure that that the timing of the LY900014 +20 arm is clearly differentiated from the premeal dosing arm. |
| Section 1. Synopsis | Updated relevant sections to match main body of protocol | |
| Section 2. Schedule of Activities | Update to footnote c | Immunogenicity follow up shortened from 1 year to 6 months based on recently obtained feedback from the FDA. |
| Section 5.1. Overall Design | Follow up for insulin lispro antibodies reduced from 48 to 26 weeks | |
| Section 5.2. Number of Participants | Increased number of participants and adjusted the screened, randomized, and completer numbers accordingly | The sample size was increased by 200 patients (100 patients for each of the double blind mealtime dosing groups) to increase the statistical power for showing superiority in HbA1c reduction between treatments at 26 weeks. |
| Section 5.3.1. Safety<br>Follow-Up | Changed Visit 805 to Visit 803 | Immunogenicity follow up shortened from 1 year to 6 months based on recently obtained feedback from the FDA. |
| Section 6.1. Inclusion<br>Criteria | Added flash glucose monitoring (FGM) | FGM is being used more commonly by patients to provide greater insight into BG profiles. Although glucose results are not provided in real time as with CGM systems, FGM can provide the patient/investigator with additional information on BG profiles that cannot be observed with SMBG alone. As with patients who use their personal CGM during the study, SMBG monitoring requirements using the study glucose meter remain the same and investigator insulin dose adjustments must be made using results from SMBG monitoring. |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Section 7.2. Method of Treatment Assignment | Replaced stratification by CGM with stratification by prandial insulin dosing plan (carbohydrate counting, pattern adjustment) | Randomization for study ITRM participants uses 4 stratification factors (country, HbA1c, basal insulin use, CGM personal use). Fewer than 10% of patients are expected to use a personal CGM or FGM system during the study. Because a potential imbalance for this factor across treatments in a small number of patients will be unlikely to influence primary objective, stratification by CGM/FGM personal use was replaced with prandial insulin dosing plan. For type 1 patients, carbohydrate counting is the preferred method for optimizing prandial insulin dose adjustment and matching insulin with carbohydrate consumption; however, pattern adjustment is still the prevailing method for prandial insulin dose adjustment used in some of the participating countries in ITRM. Given the desire to make the study applicable for management of T1D in general and to avoid mandating use of carbohydrate counting in countries where this is not the usual practice, stratification by prandial insulin adjustment method provides the best opportunity to ensure equal distribution across treatments. This resulted in a changed from a 1:1:1 randomization ratio to a 4:4:3 randomization ratio. |
| Section 7.2.1.3. Basal<br>Insulin Titration<br>Table ITRM.5 | Removed footnote a | This footnote was not consistent with the cited references and was duplicative of text appearing in the paragraph preceding Table ITRM.4 |
| Section 7.2.1.4. Study<br>Prandial Insulin<br>Therapy | Added more details on carbohydrate counting and pattern adjustment for prandial insulin dosing. Removed stratification by CGM device. | Included the option for patients who currently manage prandial insulin doses currently using the pattern adjustment method to receive training and support to learn how to use the carbohydrate counting method to determine prandial insulin dose requirements beginning at Visit 2, the start of the lead-in period. Carbohydrate counting is preferred as it provides the best option to optimize prandial insulin dose delivery with planned mealtime carbohydrate consumption. Additional guidance for transitioning onto study prandial insulin at the start of the randomization period is provided to minimize risk for postprandial hypoglycemia. |
| Section 7.3. Blinding | Added clarification | To make more specific who will remain blinded to study data |
| Section 7.6. Treatment Compliance | Added IP | To allow patients to continue study if noncompliant |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Section 9.1.4.4.<br>Mixed-Meal<br>Tolerance Test | Added more instruction | To help patients achieve the targeted fasting blood glucose level prior to start of the MMTT |
| Section 10.1. Sample<br>Size Determination | Increased sample size and updated numbers of randomized and completers | The sample size was increased by 200 patients (100 patients for each of the double blind mealtime dosing groups) to increase the statistical power for showing superiority in HbA1c reduction between treatments at 26 weeks. This resulted in a changed from a 1:1:1 randomization ratio to a 4:4:3 randomization ratio. |
| Section 10.3.1. General Statistical Considerations Section 10.3.3.1. Primary Analyses | Expanded MMRM description Replaced strata of patients personal CGM use with prandial insulin dosing plan Further explained 2 primary analysis methods; 1 for FDA submission, 1 for non-FDA submission and publication | Per request from the FDA, the primary analysis was modified for the US submission to impute missing data and use ANCOVA rather than MMRM. For other purposes, the originally planned MMRM analysis will be used. The changes in these sections reflect updates to the wording related to the primary analysis. |
| Section 10.3.3.1.1.<br>Sensitivity Analyses<br>for Missing Data | Specified ITT estimand and efficacy estimand | The strata terms in the analysis model were updated to match the changes to the stratification factors described above. |
| Section 10.3.3.1.2.<br>Additional Analyses<br>for Primary Endpoint | Deleted text | |
| Section 10.3.3.2.<br>Secondary Analyses | Added more information of graphical testing scheme Replaced strata of patients personal CGM use with prandial insulin dosing plan | |
| Section 10.3.5.2.<br>Subgroup Analyses | Added subgroup for insulin dosing plan Added FGM | |
| Section 10.3.6.<br>Interim Analyses | Added link to Section 7.3 | |

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Appendix 8 Insulin | Reduced time of follow- up to maximum of 6 | Immunogenicity follow up shortened from 1 year to 6 months based on recently |
| Lispro Antibody | months, approximately 26 weeks after Visit 801. | obtained feedback from the FDA. |
| Follow-Up | Removed Visits 804 and 805 from schedule of | |
| Assessment | activities and adjusted visit intervals to allow | |
| | antibody follow up visits 802 and 803 to occur at | |
| | approximately 3 month intervals starting from Visit | |
| | 801. | |

# **Revised Protocol Sections**

**Note:** Deletions have been identified by strikethroughs.

Additions have been identified by the use of <u>underscore</u>.

#### 1. Synopsis

#### **Objectives/Endpoints**

Multiplicity Adjusted Objectives

5. To test the hypothesis that LY900014 administered as postprandial insulin immediately after completion of a meal or at 20 minutes after the start of a meal, whichever occurs first (LY900014+20), is noninferior to insulin lispro, administered as prandial insulin, on glycemic control (NIM=0.4% for HbA1c)

#### **Treatment Groups and Duration:**

A third open-label treatment group consists of LY900014 administered immediately after completion of a meal or at 20 minutes after the start of a meal (LY900014+20), whichever occurs first.

Study visits will be scheduled at approximately 3-month intervals for up to 48-26 weeks from Visit 801 or until insulin lispro antibodies return to baseline range, whichever occurs sooner.

#### **Number of Patients:**

Approximately <u>1257-1500</u> participants will be screened to achieve <u>1005-1199</u> randomized patients and <u>852-1020</u> patients completing 26 weeks of treatment, with approximately <u>536-646</u> patients completing 52 weeks.

#### **Statistical Analysis:**

Efficacy analyses will be conducted on all randomized patients using an intention-to-treat (ITT) approach according to the treatment the patients are assigned. The analyses for the primary and multiplicity adjusted objectives will be performed for the efficacy estimand including data collected prior to permanent discontinuation of investigational product (IP) through Week 26 and for the ITT estimand (treatment regimen estimand) including all data collected through Week 26 regardless of IP use.

For the US FDA submission, the primary analysis method will use the copy reference approach to impute missing data based on multiple imputations with a pattern mixture model. This analysis is for the ITT estimand that will include all data collected from randomization through Week 26, regardless of IP use. The reference will be all observed data from the randomized patients in the same treatment arm who discontinue IP and complete the study without missing data. After imputation, the primary efficacy comparison will be based on the contrast between LY900014 and insulin lispro from the ANCOVA analysis of change from baseline to Week 26 in HbA1c using all randomized patients. The model for this analysis will include the fixed class effects of treatment and ,-strata (pooled country, type of basal insulin, and patient's personal continuous glucose monitoring [CGMprandial insulin dosing plan] use during the study), visit, and treatment by visit interaction, as well as and the continuous, fixed covariate of baseline value.

If there are only a limited number of patients in the reference group as described above that leads to a failure in performing the proposed multiple imputation analysis, the reference will be changed to include all observed data from all randomized patients in the same treatment arm who complete the study without missing data.

For non-FDA submissions and publications, the primary efficacy comparison will be based on the contrast between LY900014 and insulin lispro at Week 26 (Visit 18) from the MMRM analysis of change from baseline in HbA1c including data collected from all randomized patients prior to permanent discontinuation of IP through Week 26 (efficacy estimand). The model for this analysis will include the fixed class effects of treatment and strata (pooled country, type of basal insulin, and prandial insulin dosing plan), visit, and treatment-by-visit interaction, and the continuous, fixed covariate of baseline value.

For both primary analysis approaches, LY900014 will be declared noninferior to insulin lispro if the upper limit of the 2-sided 95% CI for the LS mean difference in the change from baseline in HbA1c for LY900014 minus insulin lispro is below +0.4%. In addition, the 95% CI for the treatment difference will be compared to an alternative NIM of +0.3%. Both estimands will be tested at the full significance level of 0.05. The ANCOVA and MMRM analyses will include data from all 3 treatment groups; however, the contrasts between LY900014+20 and insulin lispro and between LY900014 and LY900014+20 are not part of the primary efficacy comparisons.

The primary efficacy comparison will be based on the contrast between LY900014 and insulin lispro at Week 26 (Visit 18) from the mixed-effect model repeated measure (MMRM) analysis of change from baseline in HbA1e using all randomized patients. If the upper limit of the 2-sided 95% confidence interval (CI) for the least squares (LS) mean difference in the change from baseline in HbA1e for LY900014 minus insulin lispro is below +0.4%, LY900014 will be declared noninferior to insulin lispro. In addition, the 95% CI for the treatment difference from the MMRM model will be compared to an alternative NIM of +0.3%. The MMRM analysis will include data from all 3 treatment groups; however, the contrasts between LY900014+20 and insulin lispro and between LY900014 and LY900014+20 are not part of the primary efficacy comparison.

A graphical approach (Bretz et al. 2011) for multiple comparisons will be used to strongly control the overall Type I error (2-sided alpha level of 0.05) for testing the treatment effect for the primary and the following multiplicity adjusted objectives: superiority of LY900014 compared with insulin lispro for 1-hour PPG excursion at Week 26, 2-hour PPG excursion at Week 26, and change from baseline to Week 26 in HbA1c; and noninferiority of LY900014+20 to insulin lispro in change from baseline to Week 26 in HbA1c. The same graphical testing scheme will be applied for both the efficacy estimand and ITT estimand.

An analysis of covariance (ANCOVA) model with strata (pooled country, type of basal insulin, baseline HbA1c strata [(≤7.5%, >7.5%], and patient's personal CGM useprandial insulin dosing plan during the study), and treatment as fixed effects and baseline as a covariate will be used to analyze the 1-hour and 2-hour PPG excursions. However, if the percentage of the patients with missing MMTT data at baseline is higher than 15%, a constrained longitudinal data analysis model (Liu et al. 2009; Lu 2010) will be used instead. Analyses details will be documented in the statistical analysis plan (SAP).

#### 2. Schedule of Activities

Footnote c: Visit 802 should occur no sooner than approximately 9-13 weeks after Visit 801-to allow time to perform antibody testing on the Visit 801 sample.

#### 4. Objectives and Endpoints

#### **Multiplicity Adjusted Objectives**

5. To test the hypothesis that LY900014 administered as postprandial insulin immediately after completion of a meal or at 20 minutes after the start of a meal, whichever occurs first (LY900014+20), is noninferior to insulin lispro, administered as prandial insulin, on glycemic control (NIM=0.4% for HbA1c)

#### 5.1. Overall Design

A third open-label treatment group consists of LY900014 administered immediately after completion of a meal or at 20 minutes after the start of a meal (LY900014+20), whichever occurs first.

All patients who complete the 4-week safety follow-up visit (Visit 801) and have treatment-emergent insulin lispro antibodies that have not returned to the prespecified baseline range (Visit 2) will be asked to participate in follow-up to monitor insulin lispro antibody levels for up to 48 26 weeks after Visit 801 as described in Appendix 8.

At Visit 8, patients will be randomized to either LY900014 at mealtime, insulin lispro at mealtime, or LY900014 administered immediately after completion of a meal or at 20 minutes after the start of a meal (LY900014+20), whichever occurs first.

Figure ITRM. 1, footnote e Eligible patients will have visits at approximately 3-month intervals for up to 48-26 weeks after Visit 801 for follow-up of insulin lispro antibody levels (see Appendix 8).

#### 5.2. Number of Participants

Approximately 1257-1500 participants will be screened to achieve 1005-1199 randomized patients and 852-1020 patients completing 26 weeks and approximately 536-646 patients completing 52 weeks (double-blind arms only).

#### 5.3.1. Safety Follow-Up

Patients participating in the antibody follow-up period will complete the study when insulin antibodies have returned to baseline range or when Visit 805-803 is completed, whichever occurs first.

#### 5.4. Scientific Rationale for Study Design

The third treatment group is open-label due to inability to blind postprandial injection timing of LY900014 (immediately after completion of a meal or at 20 minutes after the start of a meal, whichever occurs first)

#### 6.1 Inclusion Criteria

[12] b) Perform self-BG monitoring including 10-point SMBG on designated days (patients using a personal <u>continuous glucose monitoring (CGM) or flash glucose monitoring (FGM)</u> device for insulin dosing decisions must still <del>perform the SMBG per protocol</del>use the study glucose meter according to the protocol)

#### 7.1 Treatments Administered

In a third open-label treatment group, LY900014 will be administered postprandially (immediately after completion of the meal or at 20 minutes after the start of a meal, whichever occurs first [LY900014+20]) for 26 weeks.

Table ITRM.2. Treatment Regimens

| | Dose | Dose | Route of | Timing of |
|---|---|---|---|---|
| Regimen | Strength | Administration | Administration | Administration |
| LY900014+20 | 100 U/mL | Individualized | Subcutaneous | 20 minutes after the start of the meal |
| | | dosing | | or immediately after completion of the |
| | | | | meal, whichever occurs first |

#### 7.2. Method of Treatment Assignment

Patients will be randomized to <u>double-blind LY900014</u>, <u>double-blind insulin lispro</u>, <u>or open-label LY900014+20 in a 4:4:3 ratio</u>. Stratification will be by country, HbA1c stratum (≤7.5%, >7.5% at Visit 7), type of basal insulin during the lead-in period (glargine U-100 or degludec U-100), and <u>use of patient's personal CGM systemprandial insulin dosing plan at randomization (carbohydrate counting, pattern adjustment-during the study (yes/no)</u>.

#### 7.2.1.3 Basal Insulin Titration

Table ITRM.5. Summary of Basal Insulin Adjustments after Hypoglycemia Assessment

| | When Basal Insulin ≤14 units | When Basal Insulin ≥15 units |
|---|---|---|
| If median (middle) FBG* | Adjust the basal dose by: | Adjust the basal dose by: |
| from the 3 previous FBG | | |
| values is: | | |
| ≤70 mg/dL | Decreasing dose to previous lower | Decreasing dose to previous lower |
| (≤3.9 mmol/L) | <del>dose</del> b <u>dose</u> a | <del>dose</del> b <u>dose</u> a |
| 71–100 mg/dL | No adjustment | No adjustment |
| (>3.9–5.6 mmol/L) | | |
| 101–139 mg/dL | Increasing by 1 unit | Increasing by 2 units |
| (>5.6–7.7 mmol/L) | | |
| 140–179 mg/dL | Increasing by 2 units | Increasing by 3 units |
| (>7.8–9.9 mmol/L) | | |
| ≥180 mg/dL | Increasing by 3 units | Increasing by 4 units |
| (≥10 mmol/L) | | |

Abbreviation: FBG = fasting blood glucose.

Source: Adapted from Bartley et al. 2008 and Bolli et al. 2009.

<sup>&</sup>lt;sup>a</sup> For patients using insulin glargine twice daily, investigators may also consider use of evening premeal SMBG values for assessment of morning insulin glargine dose.

ba If there is no previous dose because this was the first assigned dose after randomization, then the basal dose should be decreased by 10% in consultation with the investigator.

## 7.2.1.4. Study Prandial Insulin Therapy

Patients will be randomized (Visit 8) to either LY900014 at mealtime, insulin lispro at mealtime, or LY900014 administered immediately after completion of a meal or at-20 minutes after the start of a meal (LY900014+20), whichever occurs first.

Carbohydrate counting is the preferred method for determining prandial insulin dosing requirements. For patients entering the study using the pattern adjustment method, education and training may be provided at the start of and throughout the 8-week lead-in period to teach willing and desirous patients how to effectively use the carbohydrate counting method for determining meal time insulin doses. Patients who have demonstrated proficiency with carbohydrate counting in the opinion of the investigator should continue using this method during the treatment period.

The patient should maintain the same prandial insulin dosing plan throughout the study. <u>In order to account for potential differences between patients who manage prandial insulin doses using pattern adjustment and those who use carbohydrate counting, stratification by patients' prandial insulin dosing plan will ensure balance of this factor across treatments. -Correction factor(s) (for example, 1 unit of insulin per glucose [mg/dL or mmol/L] above target goal) may be implemented with either prandial insulin dosing plan. Adjustments in insulin dosage should also take into account conditions of stress and/or exercise and should be made individually.</u>

At randomization (Visit 8), the starting study insulin doses may be initiated unit for unit; however, investigators may consider reducing the prandial or correction insulin doses approximately 10 to-20% based on the patient's overall glycemic status or other considerations known to the investigator in order to reduce risk of postprandial hypoglycemia.

Patients who wear their personal CGM/FGM device prior to study entry will be allowed to continue to wear their CGM/FGM device during the study. However, these patients should be instructed to perform SMBG monitoring using the study glucose meter according to the protocol. In order to account for potential differences between patients who wear a CGM device and those who do not, stratification by patients' personal CGM use will ensure balance of this factor across treatments. Investigators must use the SMBG levels to make treatment decisions.

## 7.3 Blinding

A third open-label treatment group consists of LY900014 administered 20 minutes after the start of a meal (LY900014+20) , whichever occurs first.

Investigators, site staff, clinical monitors, and patients and study team members who interact directly with site personnel after primary endpoint database lock will remain blinded to the treatment assignments until the study is complete.

#### 7.6 Treatment Compliance

Patients who, in the opinion of the investigator, are deemed consistently noncompliant may be discontinued from IP or from the study.

#### 9.1.4.4. Mixed-Meal Tolerance Test

Patients should have no episodes of hypoglycemia (symptoms or BG ≤70 mg/dL [3.9 mmol/L]) during this fasting period.

**Target FBG** <u>prior to the MMTT</u>: Patients must have an FBG in the range of 71 to 180 mg/dL (3.9-10.0 mmol/L) prior to starting the MMTT. If the glucose is outside of this range, the MMTT should be rescheduled.

In order to increase the likelihood of having patients arrive on the morning of the MMTT within the target FBG range, please note the following:

- Patients should be instructed to avoid major changes in dietary intake or physical activity during the 3 days prior to the MMTT.
- Patients should be instructed to inject basal insulin according to their usual schedule
- Patients should not administer correction doses with insulin lispro or LY900014 within 4 hours of the start of the MMTT.
- During the 8 hour fasting period and up to 2 hours prior to the start of the MMTT, episodes of non-severe hypoglycemia (symptoms or BG ≤70 mg/dL [3.9 mmol/L]) can be treated with 15 to 20 grams of carbohydrate. If a hypoglycemia episode requires more than approximately 20 grams of carbohydrate within 8 hours of the start of the MMTT or the patient experiences a severe hypoglycemia episode (as defined in Sections 9.4.1 and 9.4.2), the patient should be instructed to notify the site and the MMTT must be rescheduled

## **Insulin Injection**:

Patients should inject basal insulin according to their usual schedule.

#### 10.1. Sample Size Determination

Approximately 1005-1199 patients will be randomized in order that 852-1020 patients complete the study through the primary endpoint at Week 26.

Patients will be randomized in a 1:1:14:4:3 ratio to double-blind LY900014 dosed 0 to 2 minutes before meals, double-blind insulin lispro dosed 0 to 2 minutes before meals, double-blind insulin lispro dosed 0 to 2 minutes before meals, or open-label LY900014 dosed immediately after completion of a meal or at 20 minutes after the start of a meal, whichever occurs first (LY900014+20). Assuming a noninferiority margin (NIM) of 0.4%, no true difference between treatment arms, and an SD of 1.1%, approximately 371 852 completers (284-in each double-blind treatment group) will provide at least 99% power to show noninferiority between LY900014 and insulin lispro in change from baseline to 26 weeks in HbA1c using the upper limit of a 2-sided 95% confidence interval (CI) (LY900014 – insulin lispro). Assuming a 15% dropout rate for 26 weeks, approximately 1005-1199 patients (436 in each double-blind treatment

group and 327 in the open-label treatment group) will need to be randomized. This sample size also has 9095% power to show noninferiority between LY900014 and insulin lispro using a 0.3% NIM at 26 weeks.

#### 10.3.1. General Statistical Considerations

Efficacy analyses will be conducted on all randomized patients using an intention to treat (ITT) approach-according to the treatment the patients are assigned. The analyses for the primary and multiplicity adjusted objectives will be performed for the efficacy estimand including data collected prior to permanent discontinuation of IP through Week 26 and for the ITT estimand (treatment regimen estimand) including all data collected through Week 26 regardless of IP use (Section 10.3.3.1).

The primary analysis method will be a A restricted maximum likelihood based, mixed-effect model repeated measures (MMRM) analysis using will be used to analyze continuous longitudinal variables. Aall the longitudinal observations at each scheduled postbaseline visit will be included in the analysis. The model for the analysis of the primary efficacy endpoint of change from baseline in HbA1c will include the fixed class effects of treatment, strata (pooled country, type of basal insulin, and patient's personal CGM useprandial insulin dosing plan during the study), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariate of baseline value.

An-Aanalysis of covariance (ANCOVA) will also be used to analyze continuous variables. The model for the change from baseline to the Week 26 HbA1c endpoint will include treatment and with strata (pooled country, type of basal insulin, and patient's personal-prandial insulin dosing planCGM use during the study), and treatment as fixed effects and baseline as a covariate will be conducted as supportive analyses. Unless otherwise stated, mMissing endpoints will be imputed using the last-observation—carried-forward (LOCF) approach, using only postbaseline data. For analyses of variables other than HbA1c, the HbA1c stratum ( $\leq 7.5\%$ , >7.5%) will be included in the model.

#### 10.3.3.1. Primary Analyses

The primary objective of this study is to test the hypothesis that LY900014 is noninferior to insulin lispro on glycemic control (NIM=0.4% for HbA1c) in patients with T1D, when administered as prandial insulin (0-2 minutes prior to the meal), in combination with basal insulin for 26 weeks. There will be 2 primary analysis methods, each tested at the full significance level of 0.05.

For the US FDA submission, the primary analysis method will use the copy reference approach to impute missing data based on multiple imputations with a pattern mixture model. This analysis is for The other primary estimand, requested by the US FDA, will be an the ITT estimand (effectiveness/treatment regimen estimand) that will include all data collected from randomization through Week 26, regardless of IP use. The reference will be all observed data from the randomized patients in the same treatment group who discontinue IP and complete the study without missing data. After imputation, the primary efficacy comparison will be based on

the contrast between LY900014 and insulin lispro from the ANCOVA analysis of change from baseline to Week 26 in HbA1c using all randomized patients as described in Section 10.3.1.

If there are only a limited number of patients in the reference group as described above that leads to a failure in performing the proposed multiple imputation analysis, the reference will be changed to include all observed data from all randomized patients in the same treatment arm who complete the study without missing data.

For non-FDA submissions and publications, The primary efficacy comparison will be based on the contrast between LY900014 and insulin lispro at Week 26 (Visit 18) from the MMRM analysis of change from baseline in HbA1c using including data collected from all randomized patients prior to permanent discontinuation of IP through Week 26 (efficacy estimand). If the upper limit of the 2-sided 95% CI for the LS mean difference in the change from baseline in HbA1c for LY900014 minus insulin lispro is below +0.4%, LY900014 will be declared noninferior to insulin lispro. In addition, the 95% CI for the treatment difference from the MMRM model will be compared to an alternative NIM of +0.3%. The analysis model and selection of covariance structure is described in Section 10.3.1. The MMRM analysis will include data from all 3 treatment groups; however, the contrasts between LY900014+20 and insulin lispro and between LY900014 and LY900014+20 are not part of the primary efficacy comparison.

For both primary analysis approaches, LY900014 will be declared noninferior to insulin lispro if the upper limit of the 2-sided 95% CI for the LS mean difference in the change from baseline in HbA1c for LY900014 minus insulin lispro is below +0.4%. In addition, the 95% CI for the treatment difference will be compared to an alternative NIM of +0.3%. Both estimands will be tested at the full significance level of 0.05. The ANCOVA and MMRM analyses will include data from all 3 treatment groups; however, the contrasts between LY900014+20 and insulin lispro and between LY900014 and LY900014+20 are not part of the primary efficacy comparisons.

In addition to the primary objective, the superiority of LY900014 in controlling HbA1c compared to insulin lispro will also be assessed for each analysis approach described above. If the p-value is less than the alpha level from the graphical approach allocated to the superiority hypothesis, LY900014 will be declared superior to insulin lispro.

There will be 2 primary estimands to compare treatment groups for the analysis of the primary measure of change from baseline to Week 26 in HbA1c. One primary estimand will be an efficacy estimand that includes only data collected prior to permanent discontinuation of IP through Week 26. Both estimands will use the same primary analysis model, and each will be tested at the full significance level of 0.05.

### 10.3.3.1.1. Sensitivity Analyses for Missing Data

For the ITT estimand, the reference group will be as described for the FDA primary analysis, and ANCOVA on the change from baseline to Week 26 in HbA1c will be used.

For the efficacy estimand, the reference group will be the insulin lispro treatment group. Imputation will be for all longitudinal visits.

#### 10.3.3.1.2. Additional Analyses for the Primary Endpoint

The primary MMRM analysis model, MMRM, will be repeated using the PP and Completer populations to check the sensitivity of the analysis. If the conclusion differs from that of all randomized patients, the data and analyses will be further investigated.

A secondary analysis model <u>for the efficacy estimand</u> will be an ANCOVA for HbA1c change from baseline to Week 26 (Visit 18), using the model described in Section 10.3.1. Missing endpoints will be imputed using the LOCF approach using postbaseline data only.

In addition to the primary objective, the superiority of LY900014 in controlling HbA1c compared to insulin lispro will also be assessed with the same model using all randomized patients. If the p-value is less than the alpha level from the graphical approach allocated to this hypothesis, LY900014 will be declared superior to insulin lispro.

#### 10.3.3.2. Secondary Analyses

Analyses will be performed for both the efficacy estimand and ITT estimand as described in Section 10.3.3.1 using the same graphical testing scheme.

The graphical testing scheme will be described in the SAP. The study total alpha level (or studywise type I error) is preset to be 5% for each estimand. The study total alpha level will be used for the primary objective in the initial step. The alpha level will be allocated to other key endpoints based on the weights in testing paths once the primary endpoint is successfully demonstrated. If 1 of the remaining hypotheses is successfully demonstrated with the preserved alpha level, its preserved alpha will be allocated to the remainder of the hypotheses by the weights in the paths. The iterative test procedure continues until none of the remaining hypotheses can be demonstrated with their preserved alphas or all hypotheses are demonstrated successful.

An ANCOVA model with strata (pooled country, type of basal insulin, patient's personal CGM prandial insulin dosing planuse during the study, and baseline HbA1c strata [( $\leq 7.5\%$ , >7.5%]) and treatment as fixed effects and baseline as a covariate will be used to analyze the 1-hour and 2-hour PPG excursions.

Superiority in change from baseline in HbA1c for LY900014 compared with insulin lispro and noninferiority in change from baseline in HbA1c for LY900014+20 to insulin lispro will be determined from the analysis approaches outlined in Section 10.3.3.1.

HbA1c and change from baseline in HbA1c at all time points will be analyzed by the same MMRM model used for the primary analysis for the efficacy estimand.

Additional continuous secondary efficacy variables, as well as the change from baseline for these variables, will be analyzed either by the MMRM or ANCOVA models described in Section 10.3.1 for the efficacy estimand.

Analyses of efficacy data collected from randomization through Week 52 for comparisons of the LY900014 and insulin lispro treatment groups will be similar to those described above <u>for the efficacy estimand</u>.

#### 10.3.5.2. Subgroup Analyses

- Prandial insulin dosing plan (carbohydrate counting, pattern adjustment)
- Patient's personal CGM/FGM use during the study (Yes, No)

#### 10.3.6. Interim Analyses

Investigators and patients will remain blinded to treatment assignments until the final database lock after all patients complete the study as described in Section 7.3.

#### **Appendix 8**

#### Eligibility for Insulin Lispro Antibody Follow-Up Assessment

Study visits will continue at approximately 3 month intervals for a maximum of <u>1 year6 months</u> (approximately <u>48-26</u> weeks) after Visit 801 or until insulin lispro antibodies return to baseline range, whichever occurs sooner.

Visit 802 should occur no sooner than approximately 9-13 weeks after Visit 801. to allow time to perform antibody testing on the Visit 801 sample.

In any case, even where insulin antibodies persist, the insulin lispro antibody follow-up assessment is expected to last no longer than 52-30 weeks from the protocol-scheduled last treatment visit.

#### Procedures for Insulin Lispro Antibody Follow-Up Assessment

Blood samples for insulin lispro antibody and HbA1c measurements should be collected at approximately 3-month intervals for up to 48-26 weeks after Visit 801.

Schedule of Activities during Insulin Lispro Antibody Follow-Up Assessment

| Study Period | Insulin Lispro Antibody<br>Follow-Up Period | | ED-IA<br>Follow-Up | | |
|---|---|---|---|---|---|
| eCRF Visit Number | 802 | 803 | <del>804</del> | <del>805</del> | |
| Visit Window (days) | <u>±</u> +14 | ±14 | <del>±14</del> | ±14 | |
| Time on Study Relative to Last Treatment Dose Visit (weeks) | <del>13</del> <u>17</u> | <del>26</del> 30 | <del>39</del> | <del>52</del> | |
| Time on Study Relative to First Treatment Dose Visit (weeks) | Open Label: 3943 Double Blind: 6569 | <del>52</del> <u>56</u><br><del>78</del> <u>82</u> | 65<br>91 | 7 <del>8</del> | |
| IWRS | X | X | X | X | X |
| Dispense glucose monitoring and ancillary supplies | X | X | X | | |
| Telephone call for visit reminder or informing patient of completion in the study | X | X | X | | |

| Study Period | Insulin Lispro Antibody<br>Follow-Up Period | | | | ED-IA<br>Follow-Up |
|---|---|---|---|---|---|
| eCRF Visit Number | 802 | 803 | <del>804</del> | <del>805</del> | |
| Visit Window (days) | <u>±</u> +14 | ±14 | ±14 | ±14 | |
| Time on Study Relative to Last Treatment Dose Visit (weeks) | <del>13</del> <u>17</u> | <del>26</del> <u>30</u> | <del>39</del> | <del>52</del> | |
| Time on Study Relative to First Treatment Dose Visit (weeks) | Open Label: 3943 Double Blind: 6569 | <del>52</del> <u>56</u><br><del>78</del> 82 | 65<br>91 | 78<br>104 | |
| | <del>03</del> 07 | 7002 | 71 | 107 | |
| Return of unused diabetes medications and study supplies if required by local regulations | X | X | X | X | X |
| Clinical Assessments | | | | | |
| Concomitant medication (including OAMs) | X | X | X | X | X |
| Total daily prandial insulin dose | X | X | X | X | X |
| Total daily basal insulin dose | X | X | X | X | X |
| Vital signs | X | X | X | X | X |
| Body weight | X | X | X | X | X |
| Adverse events | X | X | X | X | X |
| <b>Laboratory Assessments</b> | | | | | |
| Anti-insulin lispro antibodies | X | X | X | X | X <sup>a</sup> |
| HbA1c | X | X | X | X | X |

Leo Document ID = 1f72cd6b-be68-47a5-98a5-79f7ac33104d

Approver: PPD

Approval Date & Time: 22-May-2017 20:32:02 GMT Signature meaning: Approved

Approver: PPD
Approval Date & Time: 22-May-2017 20:39:01 GMT
Signature meaning: Approved